# **Biohaven Pharmaceuticals**

### Protocol BHV3000-303

A Phase III, Double-Blind, Randomized, Placebo-Controlled, Safety and Efficacy Trial of BHV-3000 (rimegepant) Orally Disintegrating Tablet (ODT) for the Acute Treatment of Migraine

**Statistical Analysis Plan** 

Final Version 2.0

Date: 15 November 2018

#### SIGNATURE PAGE

Protocol Title: A Phase III, Double-Blind, Randomized, Placebo-

Controlled, Safety and Efficacy Trial of BHV-3000 (rimegepant) Orally Disintegrating Tablet (ODT) for

the Acute Treatment of Migraine

Sponsor: Biohaven Pharmaceutical Holding Company Limited

Protocol Number: BHV3000-303

**Document Version/Date:** 2.0/15-November-2018

Author: PPD

# Sponsor Approval

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol, clinical development plan, and all applicable regulatory guidances and guidelines.

I have discussed any questions I have regarding the contents of this document with the biostatistical author.

I also understand that any subsequent changes to the planned statistical analyses, as described herein, may have a regulatory impact and/or result in timeline adjustments. All changes to the planned analyses will be described in the clinical study report (CSR).

| oponion or materials. | Sponsor | Signatories: |
|-----------------------|---------|--------------|
|-----------------------|---------|--------------|

PPD

# **Table of Contents**

| TABLE ( | OF CONTENTS | 3 |
|---------|-----------------------------------------------|-----|
| TABLE C | OF TABLES | 4 |
| TABLE C | OF FIGURES | 4 |
| 1 INTR | ODUCTION AND OBJECTIVES OF ANALYSIS | 8 |
| 1.1 IN | TRODUCTION | 8 |
| | UDY OBJECTIVES | |
| 1.2.1 | PRIMARY OBJECTIVES | 8 |
| 1.2.2 | SECONDARY OBJECTIVES | 8 |
| 1.2.3 | EXPLORATORY OBJECTIVES | 9 |
| 2 STUI | DY DESIGN | |
| 2.1 SY | NOPSIS OF STUDY DESIGN | .10 |
| | ANDOMIZATION METHODOLOGY | |
| 2.3 ST | UDY ESTIMANDS | .11 |
| 2.3.1 | PRIMARY ESTIMANDS | .12 |
| 2.3.2 | SECONDARY ESTIMANDS | .12 |
| 2.3.3 | EXPLORATORY ESTIMANDS | .15 |
| 3 SUBJ | ECT POPULATIONS | .16 |
| 3.1 PC | PULATION DEFINITIONS | .16 |
| | ROTOCOL DEVIATIONS | |
| 4 STAT | FISTICAL METHODS | .17 |
| 4.1 SA | MPLE SIZE JUSTIFICATION | .17 |
| 4.2 GI | ENERAL STATISTICAL METHODS AND DATA HANDLING | .18 |
| 4.2.1 | GENERAL METHODS | .18 |
| 4.2.2 | COMPUTING ENVIRONMENT | .19 |
| 4.2.3 | METHODS OF POOLING DATA | .19 |
| 4.2.4 | ADJUSTMENTS FOR COVARIATES AND STRATIFICATION | |
| 4.2.5 | MULTIPLE COMPARISONS | .19 |
| 4.2.6 | SUBPOPULATIONS | .20 |
| 4.2.7 | MISSING AND PARTIAL DATES | .22 |
| 4.2.8 | VISIT WINDOWS | .22 |
| 4.3 PL | ANNED ANALYSES | |
| 4.4 SU | BJECT DISPOSITION | .23 |
| 4.5 DF | EMOGRAPHIC AND BASELINE CHARACTERISTICS | .25 |
| | ISSING EFFICACY DATA DESCRIPTION | |
| 4.7 EF | FICACY EVALUATION | .26 |
| 4.7.1 | RESCUE MEDICATION | |
| 4.7.2 | MBS RECORDED AFTER IP IS TAKEN | |
| 4.7.3 | PRIMARY EFFICACY ENDPOINTS | .27 |
| 4.7.4 | SECONDARY EFFICACY ENDPOINTS | |
| 4.7.5 | EXPLORATORY EFFICACY ENDPOINTS | |
| 4.8 PE | IARMACOKINETIC EVALUATION | |
| | FETY EVALUATION | |
| 4.9.1 | EXTENT OF EXPOSURE | |
| 4.9.2 | ADVERSE EVENTS | |

| 4.9.3 I | ABORATORY DATA | 30 |
|---|---|---|
| 4.9.4 V | VITAL SIGNS AND PHYSICAL MEASUREMENTS | 41 |
| | CLECTROCARDIOGRAM | |
| | NON-STUDY MEDICATIONS | |
| | HEEHAN-SUICIDALITY TRACKING SCALE (S-STS) | |
| APPENDIX | | |
| APPENDIX | | |
| APPENDIX | | |
| 1 DURAL | BILITY ENDPOINTS | |
| | TAINED PAIN FREEDOM | |
| 1.2 SUS | TAINED PAIN RELIEF | 57 |
| 1.3 SUS | TAINED FREEDOM FROM MOST BOTHERSOME SYMPTOM . | 58 |
| 1.4 <b>SUS</b> | TAINED FREEDOM FROM FUNCTIONAL DISABILITY | 58 |
| | TAINED FREEDOM FROM NAUSEA | |
| 1.6 <b>SUS</b> | TAINED FREEDOM FROM PHOTOPHOBIA | 59 |
| | TAINED FREEDOM FROM PHONOPHOBIA | |
| | TO EVENT ANALYSES | |
| | E TO RESCUE MEDICATION | |
| | E TO FIRST REPORT OF ABSENCE OF VARIOUS SYMPTOMS | 61 |
| | KAPLAN-MEIER PLOTS AND TABLES: ACTUAL TIME FOR | |
| F | EVENT OF INTEREST | 62 |
| 2.2.2 F | KAPLAN-MEIER PLOTS AND TABLES: NOMINAL TIME FOR | |
| | EVENT OF INTEREST | |
| 3 PAIN A | AND MBS AT 3 HOURS POST DOSE | 62 |
| | N FREEDOM AT 3 HOURS POST DOSE | |
| | EDOM FROM MBS AT 3 HOURS POST DOSE | |
| | R ENDPOINTS AT 3 HOURS POST DOSE | |
| | EDOM FROM PHOTOPHOBIA, PHONOPHOBIA, OR NAUSEA | |
| 3 HC | OURS | 63 |
| | N RELIEF AT 3 HOURS POST DOSE | |
| | CTIONAL DISABILITY SCALE AT 3 HOURS POST DOSE | |
| APPENDIX | 4: TABLES AND FIGURES FOR SUPPORTIVE ANALYSES | 65 |
| | Toble of Tobles | |
| Table 1: | Table of Tables | 10 |
| Table 1:<br>Table 2: | Estimands for the Co-Primary Objectives | |
| | Estimands for the Secondary Objectives | |
| Table 3:<br>Table 4: | Estimands for the Exploratory Efficacy Objectives | |
| Table 4: | <b>Layout Specifications Questions Used to Determine Triptan Non-response</b> | |
| Table 5: | Evaluation Intervals for Efficacy Analysis | |
| i abic v. | Evaluation filter vals for Efficacy Alialysis | 23 |
| | Table of Figures | |
| Figure 1: | Study Schematic | 11 |
| Figure 2: | Consort Diagram | 24 |

# **ABBREVIATIONS**

| Abbreviation | Definition |
|--------------|---------------------------------------------------|
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| ASE | Asymptotic standard error |
| AST | Aspartate aminotransferase |
| AT | Aminotransferases |
| ATC | Anatomic therapeutic class |
| BOCF | Baseline observation carried forward |
| BUN | Blood urine nitrogen |
| CI | Confidence interval |
| CPK | Creatinine phosphokinase |
| CMH | Cochran-Mantel-Haenszel |
| CRF | Case report form |
| CSR | Clinical study report |
| CV | Cardiovascular |
| DILI | Drug-induced liver injury |
| ECG | Electrocardiogram |
| EDC | Electronic data capture |
| eDiary | Electronic diary |
| eDISH | Evaluation of Drug-Induced Serious Hepatotoxicity |
| eGFR | Estimated glomerular filtration rate |
| FCS | Fully conditional method |
| FDS | Functional Disability Scale |
| HDL | High-density lipoprotein |
| ICH | International Conference on Harmonization |
| IP | Investigational product |
| IRB/EC | Institutional Review Board/Ethics Committee |
| IWRS | Interactive web response system |
| LDH | Lactate dehydrogenase |
| LDL | Low-density lipoprotein |
| LOCF | Last observation carried forward |
| MBS | Most bothersome symptom |

**Abbreviation** Definition

MDRD Modification of diet in renal disease

MedDRA Medical Dictionary for Regulatory Activities

MI Multiple imputation

mITT Modified Intent-to-Treat

MQoLQ Migraine Specific Quality of Life Questionnaire

NC=F Non-Completer Equals Failure

NC1=F Non-Completer with more than 1 missing data point equals Failure

NC=M Non-Completer Equals Missing

NRS Numeric rating scale

ODT Orally Disintegrating Tablet

PID Patient identifier

POM Preference of medication

PP Per protocol set
PT Preferred term

PVD Peripheral vascular disease QD Quaque Die (one daily)

RM=F Rescue Medication = Failure

S-STS Sheehan-Suicidality Tracking Scale

SAE Serious adverse event
SAP Statistical analysis plan
SD Standard deviation

SDS Sheehan Disability Scale
SOC System Organ Class

TBL Total bilirubin

TIA Transient ischemic attack
ULN Upper limit of normal

WHO-DD World Health Organization-Drug Dictionary

### **REVISION HISTORY**

| Version | Description of Change |
|---------|-----------------------|
| 1.0 | Original Issue |

- 2.0 Add
  - Added "Revision History" table after "Abbreviations" table.
  - Section 4.7.1: Revised text for clarity and defined rescue medications.
  - Section 4.7.3.1: Added a fifth sensitivity analysis to exclude Site 002.
  - Section 4.7.3.2: Added a sixth sensitivity analysis to exclude Site 002.
  - Section 4.7.4: Specified that secondary endpoints are also assessed excluding Site 002.
  - Section 4.9.3: Specified that shift categories are independent of US and SI units, and that SI and US units are the same for ALT and AST shift categories.
  - Section 4.9.6:
    - o Changed section title to "Non-Study Medications".
    - Defined prior medications, changed definition of concomitant medications, and modified summaries of prophylactic migraine and rescue medications.

#### • Appendix 1:

- $\circ$  Modified titles of Tables 14.1.4.1 5 and Listing 16.2.2.3.
- o Renumbered 4 efficacy tables (14.2.2.7, 14.2.2.14, 14.2.2.15, 14.2.2.16)
- Added 23 tables for primary and secondary efficacy endpoints to exclude Site 002, as per changes to Sections 4.7.3.1, 4.7.3.2, and 4.7.4.
- o Removed 4 laboratory test shift tables and renumbered 4 remaining shift tables, as per changes to Section 4.9.3.
- o Added 2 tables of non-study medications, and modified the titles of the other 3 tables of non-study medications, as per changes to Section 4.9.6.

### • Appendix 3

 Section 2.2: Specified that the analysis population for functional disability was the subset of mITT subjects that reported abnormal functioning at the onset of their study migraine.

## 1 INTRODUCTION AND OBJECTIVES OF ANALYSIS

#### 1.1 Introduction

This document presents the statistical analysis plan (SAP) for Biohaven Pharmaceuticals, Protocol BHV3000-303: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Safety and Efficacy Trial of BHV-3000 (rimegepant) Orally Disintegrating Tablet (ODT) for the Acute Treatment of Migraine.

This SAP is based on the BHV3000-303, V4.0, protocol dated 23-July-2018. It contains the analysis details and methodology to answer the study objectives, including planned summary tables, by-subject listings, and figures, which will provide the basis for the results section of the clinical study report (CSR). Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analyses.

# 1.2 Study Objectives

# 1.2.1 Primary Objectives

To evaluate the efficacy of rimegepant compared with placebo in the acute treatment of migraine as measured by the co-primary endpoints of:

- Pain freedom at two hours post-dose.
- Freedom from the most bothersome symptom (MBS), associated with migraine, at two hours post-dose.

# 1.2.2 Secondary Objectives

- 1. To evaluate rimegepant compared to placebo on pain relief at 2 hours post-dose.
- 2. To evaluate the effect of rimegepant relative to placebo on the ability to function normally at 2 hours post-dose as reported on the Functional Disability scale (FDS).
- 3. To evaluate rimegepant compared to placebo on sustained pain relief from 2 to 24 hours post-dose.
- 4. To evaluate rimegepant compared to placebo on sustained freedom from MBS, associated with migraine, from 2 to 24 hours post-dose.
- 5. To evaluate rimegepant compared to placebo on the probability of requiring rescue medication within 24 hours of initial treatment.
- 6. To evaluate rimegepant compared to placebo on sustained ability to function at a normal level, as measured by the FDS, from 2 to 24 hours post-dose.

- 7. To evaluate rimegepant compared to placebo on sustained pain relief from 2 to 48 hours post-dose.
- 8. To evaluate rimegepant compared to placebo on freedom from the MBS, associated with migraine, from 2 to 48 hours post-dose.
- 9. To evaluate rimegepant compared to placebo on the sustained ability to function at a normal level, as measured by the FDS, from 2 to 48 hours post-dose.
- 10. To evaluate rimegepant compared to placebo on freedom from photophobia at 2 hours post-dose.
- 11. To evaluate the effect of rimegepant relative to placebo on the ability to function at a "normal" level at 90 minutes post-dose as reported on the FDS.
- 12. To evaluate rimegepant compared to placebo on pain relief at 90 minutes post-dose.
- 13. To evaluate rimegepant compared to placebo on sustained pain freedom from 2 to 24 hours post-dose.
- 14. To evaluate rimegepant compared to placebo on freedom from the MBS, associated with migraine, at 90 minutes post-dose.
- 15. To evaluate rimegepant compared to placebo on pain freedom at 90 minutes post-dose.
- 16. To evaluate rimegepant compared to placebo on freedom from phonophobia at 2 hours post-dose.
- 17. To evaluate rimegepant compared to placebo on sustained pain freedom from 2 to 48 hours post-dose.
- 18. To evaluate rimegepant compared to placebo on pain relief at 60 minutes post-dose.
- 19. To evaluate the effect of rimegepant relative to placebo on the ability to function at a "normal" level at 60 minutes post-dose, as reported on the FDS.
- 20. To evaluate rimegepant compared to placebo on freedom from nausea at 2 hours post-dose.
- 21. To evaluate rimegepant compared to placebo for the incidence of pain relapse from 2 to 48 hours post-dose.

# 1.2.3 Exploratory Objectives

1. To evaluate the effect of rimegepant relative to placebo on the subjects' ability to work or function at 24 hours post-dose according to the FDS.

- 2. To evaluate the effect of rimegepant compared to placebo on pain relief at 30 minutes post-dose.
- 3. To evaluate the effect of rimegepant compared to placebo on pain relief at 15 minutes post-dose.
- 4. To evaluate the effect of rimegepant relative to placebo on the Migraine Preference of Medication (PoM).
- 5. To evaluate rimegepant relative to placebo for pain relief on the 4-point scale at all scheduled time points post-dose.
- 6. To evaluate the effect of rimegepant relative to placebo on the Migraine Quality of Life Questionnaire (MQoLQ).
- 7. To evaluate the tolerability and safety of rimegepant in the acute treatment of migraine as measured by the frequency of adverse events of at least moderate intensity, serious adverse events, and clinically relevant laboratory abnormalities.
- 8. To evaluate the effect of rimegepant (75 mg ODT) relative to placebo on the Sheehan Suicidality Tracking Scale (S-STS).

# 2 STUDY DESIGN

# 2.1 Synopsis of Study Design

BHV3000-303 is a Phase III, multicenter, randomized, double-blind, 2-arm placebo-controlled parallel-group study designed to assess safety and efficacy in the treatment of moderate to severe migraine.

After providing informed consent, subjects will first participate in the screening phase (3-28 day period) to determine eligibility for the study.

After randomization, the subject will be dispensed a single dose of the double-blind study medication consisting of a rimegepant 75 mg ODT (administered sublingually) or matching placebo to take home for up to 45 days. This study medication is to be taken when a migraine attack reaches moderate or severe intensity on the numeric rating scale (NRS) as indicated in the electronic diary (eDiary). The subject will complete an eDiary for up to 48 hours after taking the study medication. Subjects will record efficacy data in their eDiary and will telephone the study center immediately if a severe or serious adverse event occurs.

Subjects will return to the study site within 7 days of study treatment for review of the eDiary, assessment of medication compliance, and monitoring of tolerability and safety. If a subject has NOT experienced a migraine headache of sufficient severity within the 45 days after randomization, they still are required to complete all EOT visit procedures and return unused study medication and eDiary to the study center.

# 2.2 Randomization Methodology

Subjects in this study may be randomized only once. Under no circumstances may a subject be re-randomized.

The study will randomize approximately 1,430 subjects. The subjects will be randomized in a 1:1 ratio to receive rimegepant in a 75 mg ODT or matching placebo (see Figure 1). The randomization will be stratified by the use of prophylactic migraine medications (yes or no).

Figure 1: Study Schematic



# 2.3 Study Estimands

The tables that follow lay out the estimands corresponding to the study objectives. In these tables, the following abbreviations are used to describe the handling of intercurrent events for efficacy estimands:

#### **NC=F:** Non-Completers = Failure.

A subject with any missing data for an endpoint is classified as a treatment failure.

#### NC1=F: Non-Completers with more than 1 missing data point = Failure.

Subjects with more than 1 missing data point, other than at the 2, 24 or 48 hour data points, are classified as treatment failures. This applies to endpoints that are based on data from multiple time points. For example, for the durability endpoint of sustained pain freedom from 2 to 24 hours, the subjects should provide data at 2, 3, 4, 6, 8, and 24 hours. For NC1=F imputation, the data at 2 and 24 hour time points must be present or the subject is classified as a failure. However, any single data point may be missing at 3, 4, 6 or 8 hours without penalty. For

sustained pain freedom from 2 to 48 hours, the data at 2, 24, and 48 hours are required to be present.

#### **RM=F:** Rescue Medication = Failure.

Subjects that take rescue medication before, or at, the time of the event of interest are classified as failures. If the time of rescue medication is missing, all events on or after the date of rescue medication are classified as failures.

## 2.3.1 Primary Estimands

The estimands corresponding to the co-primary objectives for this study are shown in Table 1.

The population summary for all primary estimands is the difference in the percentage of subjects with a positive result ('risk difference') between the BHV-3000 and the Placebo treatment groups. This summary is computed using the modified Intent-to-Treat (mITT) population as defined in section 3.1.

Table 1: Estimands for the Co-Primary Objectives

| Objective | Pain Freedom at 2 hours post-dose |
|---|---|
| Population | mITT |
| Variable | Percent of subjects reporting no pain at 2 hours post-dose |
| <b>Intercurrent Events</b> | NC=F; RM=F. |
| Objective | Freedom from Most Bothersome Symptom (MBS) |
| Population | mITT |
| Variable | Percent of subjects reporting absence of their MBS at 2 hours post dose |
| Intercurrent Events | NC=F; RM=F; Failure to report MBS = F; Study medication taken before reporting MBS=F. |

# 2.3.2 Secondary Estimands

The estimands corresponding to the secondary objectives are shown in Table 2.

The population summary for all secondary estimands is the difference in the percentage of subjects with a positive result ('risk difference') between the BHV-3000 and the Placebo treatment groups.

# Table 2: Estimands for the Secondary Objectives

| Objective | Dain Daliaf (at 60 minutes 00 minutes or 2 hours) |
|---|---|
| • | Pain Relief (at 60 minutes, 90 minutes, or 2 hours) mITT |
| Population<br>Variable | |
| | Percent of subjects who report mild or no pain at the specified timepoint |
| Intercurrent Events | NC=F; RM=F |
| Objective | Functional Disability (at 60 minutes, 90 minutes, or 2 hours) |
| Population | mITT |
| Variable | Percent of subjects with a response of "normal" at the specified timepoint |
| Intercurrent Events | NC=F; RM=F |
| Objective | Sustained Pain Relief (2 to 24 hours; or 2 to 48 hours) |
| Population | mITT |
| Variable | Percent of subjects who report no pain or mild pain during the period of interest |
| Intercurrent Events | NC1=F; RM=F |
| Objective | Sustained Freedom from MBS (2 to 24 hours; or 2 to 48 hours) |
| Population | mITT |
| Variable | Percent of subjects who report freedom from MBS during the period of interest |
| Intercurrent Events | NC1=F; RM=F |
| Objective | Probability of Rescue Medication within 24 hours post-dose |
| Population | mITT |
| Variable | Percent of subjects taking rescue medication within 24 hours post-dose |
| Intercurrent Events | None |
| Objective | Sustained Normal Functioning (2 to 24 hours; or 2 to 48 hours) |
| Population | mITT |
| Variable | Percent of subjects who report normal functioning on the FDS during the period of |
| | interest |
| Intercurrent Events | NC1=F; RM=F |
| Objective | Photophobia Freedom at 2 hours post-dose |
| Population | mITT subjects with photophobia reported as present at migraine onset |
| Variable | Percent of subjects reporting no photophobia at 2 hours post-dose |
| Intercurrent Events | NC=F; RM=F |
| Objective | Sustained Pain Freedom (2 to 24 hours; or 2 to 48 hours) |
| Population | mITT |
| Variable | Percent of subjects who report no pain during the period of interest |
| Intercurrent Events | NC1=F; RM=F |
| Objective | MBS Freedom at 90 minutes post-dose |
| Population | mITT subjects |
| Variable | Percent of subjects reporting freedom from MBS at 90 minutes post-dose |
| Intercurrent Events | NC=F; RM=F |
| Objective | Pain Freedom at 90 minutes post-dose |
| Population | mITT |
| Variable | Percent of subjects who report no pain at 90 minutes post-dose |
| Intercurrent Events | NC=F; RM=F |
| Objective | Phonophobia Freedom at 2 hours post-dose |
| Population | mITT subjects with phonophobia reported as present at migraine onset |
| Variable | Percent of subjects reporting no phonophobia at 2 hours post-dose |
| Intercurrent Events | NC=F; RM=F |
| Intercurrent Events | 110 1, 1011 1 |

| Objective | Nausea Freedom at 2 hours post-dose |
|---|---|
| Population | mITT subjects with nausea reported as present at migraine onset |
| Variable | Percent of subjects reporting no nausea at 2 hours post-dose |
| Intercurrent Events | NC=F; RM=F |
| Objective | Pain Relapse (2 to 48 hours) |
| Population | mITT subjects who report pain freedom at 2 hours post-dose |
| Variable | Percent of subjects who report any pain during the period of interest |
| Intercurrent Events | NC1=F; RM=F |

# 2.3.3 Exploratory Estimands

The estimands corresponding to the exploratory objectives are shown in Table 3.

**Table 3: Estimands for the Exploratory Efficacy Objectives** 

| Objective | Functional Disability at 24 hours |
|---|---|
| Population | mITT |
| Variable | Percent of subjects with a response of "normal" at 24 hours post-dose |
| <b>Intercurrent Events</b> | NC=F; RM=F |
| Pop. Summary | Percentage within each treatment group (BHV3000 & Placebo) |
| Objectives | Pain Relief at 15 and 30 minutes post-dose |
| Population | mITT |
| Variable | Percent of subjects who report pain as mild or none at the time point of interest |
| <b>Intercurrent Events</b> | NC=F; RM=F |
| Pop. Summary | Percentage within each treatment group (BHV3000 & Placebo) |
| Objectives | Preference of Medication |
| Population | Treated subjects who: 1) answer "yes" to the lead-in question (i.e. "Have you ever taken migraine medication?") and provide preference of medication data |
| Variable | Percentage of subjects who prefer study medication to previous migraine medications |
| <b>Intercurrent Events</b> | Observed analysis. No accounting for intercurrent events. |
| Pop. Summary | Percentage within each treatment group (BHV3000 & Placebo) |
| Objectives | Pain Relief, on a 4 point scale, at all time points |
| Population | mITT |
| Variable | Percent of subjects who report pain as none, mild, moderate or severe |
| Intercurrent Events | NC=F; RM=F |
| Pop. Summary | Percentage of each response, in each treatment group (BHV3000 & Placebo) |
| Objectives | Migraine Quality of Life Questionnaire |
| Population | mITT |
| Variable | Total score on the MQoLQ |
| <b>Intercurrent Events</b> | Observed analysis. No accounting for intercurrent events. |
| Pop. Summary | Average total score within each treatment group (BHV3000 & Placebo) |
| Objective | Safety and Tolerability |
| Population | All treated subjects |
| Variables | Multiple |
| Intercurrent Events | Subjects analyzed as treated. No accounting for intercurrent events |
| Pop. Summary | Multiple (discussed under section 6, "Safety Analyses") |
| Objective | Sheehan Suicidality Tracking Scale |
| Population | All treated subjects |
| Variables | Change from baseline in the total score |
| <b>Intercurrent Events</b> | Subjects analyzed as treated. No accounting for intercurrent events |
| Pop. Summary | Percentage of subjects, by treatment group, in each of 5 categories (<-1, -1, no change, 1, >1) |

### 3 SUBJECT POPULATIONS

# 3.1 Population Definitions

The following subject populations will be evaluated and used for presentation and analysis of the data:

Enrolled subjects: subjects who sign an informed consent form and are assigned a subject identification number.

Randomized subjects: enrolled subjects who receive a randomization treatment assignment from the interactive web response system (IWRS).

Treated subjects: enrolled subjects who take any amount of study therapy (rimegepant or placebo).

Modified Intent-to-Treat (mITT) subjects: enrolled subjects who are randomized only once, take study therapy, have a baseline migraine of moderate to severe intensity, and who provide at least one post-baseline efficacy data point.

#### 3.2 Protocol Deviations

A protocol deviation is any variance from the approved protocol, either intentional or unintentional. The possible categories for all protocol deviations are as follows:

- Informed Consent
- Inclusion/Exclusion Criteria (specify #)
- Concomitant Medication
- Serious Adverse Event (SAE) Reporting
- Regulatory
- Drug Storage/Preparation
- Drug Administration
- Visit Schedule
- EPro Diary Noncompliance
- Noncompliance (i.e., trends, missed assessments).

A significant protocol deviation is any deviation that could impact subject safety or the integrity of the trial. For the purposes of this study, significant protocol deviations will be defined as the following:

- Inadequate informed consent or initiation of study procedures prior to completing the informed consent
- Enrollment of subjects not meeting the inclusion/exclusion criteria
- Unreported SAEs
- Improper breaking of the blinding of the study
- Use of prohibited medication as defined by the protocol
- eDiary non-compliance with primary and secondary endpoints (2, 24, or 48-hour post-dose assessment
- Repeated deviations of the same nature for a given site or subject
- Initiation of rescue medication(s) prior to primary endpoint at 2-hours

The sponsor, or designee, will be responsible for producing the final protocol deviation file (formatted as a Microsoft Excel file). This file will include site, subject ID, deviation date, deviation type, and a description of the protocol deviation.

All protocol deviations (with the exception of those related to rescue medication and missed eDiary assessments) will be presented in a by-subject listing. Handling of rescue medication and missed eDiary assessments are described in the statistical methods section of this SAP.

### 4 STATISTICAL METHODS

## 4.1 Sample Size Justification

If roughly 85% of the 715 subjects randomized to each treatment arm have a migraine in the allotted time period, there will be approximately 600 treated subjects per group.

Based on data from studies BHV3000-301 and BHV3000-302, 600 treated subjects per arm provides 95% power to detect a difference between rimegepant and placebo on the subject's self-reported most bothersome symptom. Also, 600 subjects per arm provides 95% power to detect a difference in freedom from pain at 2 hours post dose. Having 95% power on each coprimary endpoint provides roughly 90% power to detect a difference on both endpoints jointly.

# 4.2 General Statistical Methods and Data Handling

## 4.2.1 General Methods

All output will be incorporated into Microsoft Excel or Word files, sorted and labeled according to the International Conference on Harmonization (ICH) recommendations, and formatted to the appropriate page size(s). PDF versions of the output will also be produced.

Tabulations will be produced for appropriate demographic, baseline, efficacy, safety, and other parameters by as-randomized treatment group (BHV3000, Placebo) and overall, unless specified otherwise. For categorical variables, summary tabulations of the number and percentage of subjects within each category will be presented. If applicable, a category for missing data will also be presented. For continuous variables, descriptive statistics (e.g., n, mean, median, SD, minimum, and maximum) will be presented. The minimum and maximum will be presented with the same precision as the data. The mean and median will be presented with the precision of the data + 1 decimal place. The SD will be presented with the precision of the data + 2 decimal places.

Formal statistical hypothesis testing and summary statistics will be presented, as well as confidence intervals (CIs) on selected endpoints, as described in the sections below.

The default tables, listings, and figures layout will be as presented in Table 4 below:

Table 4: Layout Specifications

| Orientation | Portrait | Landscape |
|---|---|---|
| Paper Size | Letter | Letter |
| Margins | Top: 3.05 cm<br>Bottom: 2.54 cm<br>Left: 2.54 cm<br>Right: 2.54 cm | Top: 3.05 cm<br>Bottom: 2.2 cm<br>Left: 1.9 cm<br>Right: 1.9 cm |
| Font | Table text: Times new Roman<br>9 or 10 pts<br>Table title: Times new Roman<br>12 pts<br>Table legend: Times new<br>Roman 10 pts | Table text: Times new Roman<br>8, 9 or 10 pts<br>Table title: Times new Roman<br>12 pts<br>Table legend: Times new<br>Roman 9 or 10 pts |

The font size may be reduced as necessary to allow additional columns to be presented, but not at the expense of clarity. Also the orientation may be changed to portrait if appropriate.

Unless specified otherwise, by-subject listings will be sorted by site, subject ID, and additional variables such as time points, as applicable. Listings will display site-subject ID and asrandomized treatment group (as-treated treatment group for safety).

# 4.2.2 Computing Environment

All statistical analyses will be performed using SAS statistical software (Version 9.4). Medical history and adverse events (AEs) will be coded using the latest available version of Medical Dictionary for Regulatory Activities (MedDRA). Concomitant medications will be coded using the latest available version of World Health Organization Drug Dictionary (WHO-DD).

## 4.2.3 Methods of Pooling Data

In the case of sparse data for the stratification factor (use of prophylactic medication: yes or no), the responses will be pooled in summary tables. Specific details on the procedures for pooling data are presented in the applicable sections of the document outlining the analyses.

# 4.2.4 Adjustments for Covariates and Stratification

The randomization of subjects is stratified by the use of prophylactic migraine medication (yes or no). Hence, most analyses are stratified by the use or prophylactic medication.

## 4.2.5 Multiple Comparisons

Type I error is controlled in this study by using a hierarchical gate-keeping procedure. First, the family of two co-primary endpoints is tested. If the co-primary endpoints are both found to be significant, then secondary endpoints are tested in a fixed sequence. In particular, each co-primary endpoint will be tested for superiority to placebo at a two-sided alpha level of 0.05 without further adjustment for multiplicity. If the primary endpoint tests are both significant, then the following secondary endpoints will be tested in a fixed sequence, in the order shown, with each test conducted at p=0.05:

- 1. Pain Relief at 2 hours
- 2. Functional Disability at 2 hours
- 3. Sustained Pain Relief from 2 to 24 hours
- 4. Sustained Freedom from MBS from 2 to 24 hours
- 5. Probability of Rescue Medication within 24 hours
- 6. Sustained Normal Functioning (on FDS) from 2 to 24 hours
- 7. Sustained Pain Relief from 2 to 48 hours
- 8. Sustained Freedom from MBS from 2 to 48 hours
- 9. Sustained Normal Functioning (on FDS) from 2 to 48 hours
- 10. Freedom from Photophobia at 2 hours

- 11. Functional Disability at 90 minutes
- 12. Pain Relief at 90 minutes
- 13. Sustained Pain Freedom from 2 to 24 hours
- 14. MBS Freedom at 90 minutes
- 15. Pain Freedom at 90 minutes
- 16. Freedom from Phonophobia at 2 hours
- 17. Sustained Pain Freedom from 2 to 48 hours
- 18. Pain Relief at 60 minutes
- 19. Functional Disability at 60 minutes
- 20. Freedom from Nausea at 2 hours
- 21. Pain Relapse from 2 to 48 hours

If a test in the hierarchy is not significant, then any further tests on endpoints in the sequence will have p-values presented only for descriptive purposes, and no conclusions will be drawn from those results.

For exploratory endpoints, no attempt will be made to adjust for multiplicity. Any exploratory endpoints for which p-values are produced will be evaluated at an unadjusted two-sided alpha level of 0.05 and presented only for descriptive purposes.

# 4.2.6 Subpopulations

The subgroups of interest for this study:

Age: Categorized as  $< 40, \ge 40$  years

Race: white, black or African American, other (including Asian), Asian only. Certain tables may be created for the Asian population only; but in the subgroup analyses, Asian subjects will generally be included in the "other" category due to low counts.

Sex: Female/Male

Aura: Presence/Absence

Headaches per Month: Categorized as < median, ≥ median, where median is calculated overall across treatment groups combined for mITT subjects.

Triptan Non-Responder: Yes/No

Cardiovascular (CV) Risk Contraindicating Triptans: Yes/No

Subgroup analyses will be performed for the primary efficacy endpoints only.

Triptan non-responders are identified using the "Prior Triptan Response" Case Report Form (CRF) pages, which capture reasons for discontinuing triptans taken historically. The definition of triptan non-responder is based on the number of triptans that a subject failed for efficacy reasons. For each triptan and route of administration, the subject is asked the questions shown in Table 5. A subject is considered to have failed a drug for efficacy reasons if they indicated "most or all of the time" for any of the reasons in the table.

A triptan non-responder is defined as any subject that fails two or more molecular entities for efficacy reasons. To be considered a failure for a molecular entity, the subject must have failed on all routes of administration that the subject tried for the molecular entity.

Table 5: Questions Used to Determine Triptan Non-response

| | Most or All of the Time | Some of the Time | Rarely | Never |
|---|---|---|---|---|
| The treatment took too long to relieve my headache pain. | | | | |
| The pain returned after it was relieved within 24 hours | | | | |
| The treatment did not relieve my other symptoms (nausea, sensitivity to light or sound, for example). | | | | |
| I could not count on this treatment to relieve<br>my pain and symptoms every time | | | | |

Subjects with CV risk that contraindicates triptans are identified using the "Cardiac and Other Risk Factors" CRF pages. The pages are used to identify subjects with cardiovascular conditions cited in triptan labels as contraindications. A subject is identified as someone with cardiovascular risk factors contraindicating triptans if any of the following questions are answered as "yes":

Does the subject have ischemic coronary artery disease?

Does the subject have coronary artery vasospasm including Prinzmetal's angina?

Does the subject have Wolff-Parkinson-White Syndrome or arrhythmias associated with other cardiac accessory conduction pathway disorders?

Does the subject have history of stroke or transient ischemic attack (TIA)?

Does the subject have peripheral vascular disease (PVD)?

Does the subject have ischemic bowel disease?

Does the subject have uncontrolled hypertension?

# 4.2.7 Missing and Partial Dates

For efficacy analyses, partial or missing dates will not be imputed. The relative study days, where determined, will be calculated for full dates only.

For rescue medication, if the time of rescue medication is missing, then all endpoints on or after the date of rescue medication will be imputed as failures.

For missing and/or partial dates regarding non-study medications, a conservative approach will be taken. The medication will be assumed to be concomitant if it cannot be definitively shown that the medication was not taken after the period beginning 14 days prior to the taking of study medication.

If the start date of an AE is partially or completely missing, then the date will be compared as far as possible with the date of the randomization. The AE will be assumed to be on-study if it cannot be definitively shown that the AE did not occur or worsen during the post-randomization period (worst case approach).

The following general rules will be used:

If the start day is missing, but the start month and year are complete, an AE will only be excluded as being on-study if the start month/year is before the month/year of randomization or if the stop date is before randomization.

If the start day and month are missing, but the start year is complete, an AE will only be excluded as being on-study if start year is before the year of randomization or if the stop date is before randomization.

If the start date is completely missing, an AE will be considered on-study unless the stop date is before randomization.

#### 4.2.8 Visit Windows

Windows for the timeframe around efficacy measurements (15, 30, 45, 60, 90 minutes, 2, 3, 4, 6, 8, 24, and 48 hours) will be automated and captured in the eDiary. Refer to Table 6 for details on the evaluation intervals and Appendix 2 for details on the schedule of assessments.

Table 6: Evaluation Intervals for Efficacy Analysis

| Evaluation | Protocol-Specified Interval | Analysis-Specified Interval |
|---|---|---|
| Screening Phase | | |
| Screening | Day -28 to Day -3 | Day -40 to Day -3 |
| Acute (Randomization) Phase | | |
| Baseline (Randomization) | Day 1 | Day -2 to 1 |
| Onset of Migraine | Day 1 to 45 | Day 1 to 45 |
| 15, 30, 45, 60, 90 minutes post-<br>dose | Time of Dose + 15, 30, 45, 60, and 90 minutes | Time of Dose + 15, 30, 45, 60, and 90 minutes (as captured in eDiary) |
| 2 hours post-dose | Time of Dose + 2 hours | Time of Dose + 2 hours (as captured in eDiary) |
| 3 hours post-dose | Time of Dose + 3 hours | Time of Dose + 3 hours (as captured in eDiary) |
| 4 hours post-dose | Time of Dose + 4 hours | Time of Dose + 4 hours (as captured in eDiary) |
| 6 hours post-dose | Time of Dose + 6 hours | Time of Dose + 6 hours (as captured in eDiary) |
| 8 hours post-dose | Time of Dose + 8 hours | Time of Dose + 8 hours (as captured in eDiary) |
| 24 hours post-dose | Time of Dose + 24 hours | Time of Dose + 24 hours (as captured in eDiary) |
| 48 hours post-dose | Time of Dose + 48 hours | Time of Dose + 48 hours (as captured in eDiary) |
| End of Treatment Visit | Time of Dose + 7 days | > Day of Dose + 2 days (as defined by visit) |

## 4.3 Planned Analyses

Study Day 1 is defined as the day of randomization. The analyses planned for endpoints that use data from this study only will be conducted after the last subject completes their End of Treatment Visit or discontinues from the study, and the database has been locked.

# 4.4 Subject Disposition

A summary of subject disposition will be tabulated for all enrolled subjects by treatment group and overall. The disposition table will support the creation of a consort diagram, similar to that shown in Figure 1. The categories in the table will include:

Number of subjects screened

Number of screened subjects excluded from the study and reason for exclusion

Number of subjects randomized

Number of subjects not treated, and the reasons for not being treated

Number of subjects treated, and their status

Completed Study

Discontinued, and reasons for discontinuation

Number of subjects in each analysis population

A by-subject listing of subject disposition information, including the reason for discontinuation, if applicable, will be presented.

Figure 2: Consort Diagram



# 4.5 Demographic and Baseline Characteristics

Demographic information, medical history by system organ class (SOC) and preferred term (PT), migraine history, cardiovascular risk factors, and prior/current triptan response will be summarized by as-randomized treatment group and overall for the mITT population to support efficacy. A similar set of tables will be made for the treated population by as-treated treatment group and overall to support safety.

A separate set of tabulations, including demographic information and migraine history, will be made for subjects enrolled but not randomized (overall only) and subjects randomized but not treated (by as-randomized treatment group and overall).

Demographic and other baseline data will also be provided in by-subject data listings.

For each subject, multiple medical histories of the same SOC or PT will be counted only once within each SOC and PT. Medical histories will be presented in descending order of overall frequency within SOC and PT.

# 4.6 Missing Efficacy Data Description

Descriptions and tabulations of missing data will only be concerned with the post-baseline time points required for computation of the primary and secondary endpoints, and will be assessed as-randomized. These include the time points measured from 2 hours through 48 hours post-dose (e.g.: 60 minutes, 90 minutes, 2, 3, 4, 6, 8, 24 and 48 hours). The other time points (15, 30, 45 minutes) are only required for the exploratory endpoints. Also, some tabulations focus on the pain endpoint as that should be generally descriptive of the other efficacy endpoints.

The number and percentage of (1) randomized subjects who do not meet the criteria for the mITT population, and (2) randomized and treated subjects who do not meet the criteria for the mITT population will be tabulated by treatment group and overall.

For the mITT population, the items below will be tabulated by treatment group and overall.

Number and percentage of subjects with missing pain data at each time point from 2 through 48 hours post-dose. The categories in this tabulation are not mutually exclusive as subjects may have missing data at multiple time points.

Number and percentage of subjects with: no missing pain data; 1 missing time point, 2 missing time points, 3 missing time points, 4 missing time points, 5 missing time points, 6 missing time points, or 7 missing time points. The categories in this tabulation are mutually exclusive.

The number and percentage of subjects with missing data on the following endpoints measured at 2-hours post-dose: pain, MBS, photophobia, phonophobia, nausea, and functional disability.

In addition, the number and percentage of mITT subjects with missing pain data at 2 hours post-dose will be displayed by treatment group and overall within the categories of each of the following subgroups:

Age: Categorized as < 40 or  $\ge 40$  years

Race: white; black or African American; other (including Asian); Asian only

Sex: Female or Male

Aura for study migraine: Presence or Absence

Headaches per Month: Categorized as < median or  $\ge$  median (see Section 4.2.6)

Triptan Non-Responder: Yes/No

Rescue medication taken at any time during the study: Yes/No

MBS at migraine onset: photophobia, phonophobia, nausea, and not reported

# 4.7 Efficacy Evaluation

Unless otherwise noted, all efficacy analyses will be conducted using the mITT population as outlined below. Efficacy tabulations will present results by as-randomized treatment group only (excluding overall), unless specified otherwise. All efficacy data will be included in listings by subject, treatment group, and time point (as applicable).

For efficacy analyses, baseline is considered as the assessment at the onset of the treated migraine.

#### 4.7.1 Rescue Medication

Subjects who take rescue medication will be considered as failures for any efficacy evaluations that are on or after the first rescue medication date/time. If the time of first rescue medication is missing, subjects will be considered as failures for any efficacy evaluations that are on or after the first rescue medication date.

Rescue medications are defined as non-study medications reported on the Rescue Medication CRF with complete medication dates, and either (1) medication date/time after the study drug first dose date/time, or (2) medication date equal to study drug first dose date if the medication time is missing.

The first rescue medication date/time is defined as the earliest rescue medication date/time, where missing time is considered to be earlier than non-missing time on the same date.

#### 4.7.2 MBS Recorded After IP is Taken

Subjects that record their MBS after taking the investigational product (IP) are considered failures for the analysis of MBS.

# 4.7.3 Primary Efficacy Endpoints

In addition to the analyses described below, data regarding the co-primary efficacy endpoints, pain freedom and freedom from MBS at 2 hours post-dose will be presented in a by-subject listing that includes treatment group, historical MBS, MBS at time of onset of study migraine, initial migraine severity, gender, presence or absence of aura, and use of prophylactic migraine medication.

#### 4.7.3.1 Pain Freedom at 2 Hours Post-Dose

Pain freedom is assessed using the number of mITT subjects that report pain levels of "none" at 2 hours post-dose on a 4-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe). The information from the 4-point scale is directly summarized as follows:

A table showing descriptive statistics for the observed data, which includes the number and percentage of subjects reporting each of the 4 pain levels at 2 hours post-dose, and the percentage of subjects with missing data, for each treatment group. The table will include exact (Clopper-Pearson) 95% CIs for each percentage. This table will be repeated for Asian subjects only.

The estimand for the primary analysis is the percentage of pain free subjects. In statistical terms, this percentage is arrived at by estimating the probability or the "risk" that a subject is pain free.

The population summary, the between group difference in the percentage of pain free subjects is assessed by computing the "risk difference" between treatment groups. This is evaluated by computing the common risk difference, using Cochran-Mantel-Haenszel (CMH) weights (sample size weights), stratified by the use of prophylactic migraine medication (yes or no). The risk difference is tested at a two-sided alpha level of 0.05. Missing data at 2 hours post-dose will be imputed as failures (NC=F). If a stratum (prophylactic medication use: yes or no) has sparse data (less than 5 subjects), then the strata will be pooled.

Results presented for the primary analysis include the following:

- The number and percentage of subjects who are pain free, and those not pain free, at 2 hours post-dose. These are presented by stratum and treatment group, with asymptotic standard errors (ASE), and 95% asymptotic CIs.
- Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.
- Risk difference within each stratum with sample size, p-value, ASE, and 95% asymptotic CIs.

- A forest plot of the risk differences within each stratum, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

The primary analysis will be repeated for the subgroups described in Section 4.2.6.

Sensitivity analyses will be conducted as follows:

- 1. The primary analysis is repeated, using the mITT population, with missing data at 2 hours post-dose imputed using Last Observation Carried Forward (LOCF). Baseline Observation Carried Forward (BOCF) is permitted.
- 2. The primary analysis is repeated using only data from complete cases (data present at baseline and 2 hours).
- 3. The primary analysis is executed using the mITT population, and multiple imputation (with 20 imputations; m=20) methods to impute missing data at 2 hours post-dose using the copy from reference approach. The fully conditional specification (FCS) method is used with a generalized logit distribution. Covariates may include use of prophylactic medication (yes or no), sex, migraine intensity at onset (severe or other), migraines per month (< median, ≥ median), and the subject's MBS at time of study migraine onset (nausea, photophobia, or phonophobia).
- 4. A series of "what if" analyses are conducted that show what the analysis results would look like if the missing data in each treatment group were replaced with data from subjects having success rates that vary over the range of 0, 10, 20 and 30 percent. The results of this analysis are presented in a 4x4 matrix, with the rows representing the success rates for the placebo group and the columns representing the success rates for the BHV-3000 group. For example, the "30,0" cell shows the hypothetical result when a responder rate of 30% replaces the missing placebo data, and a responder rate of 0% replaces the missing BHV-3000 data. Each cell in this table will show the common risk difference, asymptotic 95% CI and uncorrected p-value. The table will be accompanied by a forest plot that displays the 16 CIs.

## 4.7.3.2 Freedom from MBS at 2 Hours Post-Dose

Freedom from each subject's MBS is assessed using the number of mITT subjects who report that their MBS (reported at migraine onset) is absent at 2 hours post-dose. The symptoms that can be nominated as the MBS (phonophobia, photophobia or nausea) are measured using a binary scale (0=absent, 1=present).

Subjects who reported their MBS after taking IP, or who did not provide an MBS are considered failures in this analysis.

Tabulations will be presented as follows:

The number and percentage of subjects reporting each of the migraine associated symptoms (phonophobia, photophobia or nausea) by treatment group and overall as most bothersome, subjects with a missing MBS, and subjects who reported their MBS after taking study medication.

An overall cross tabulation of the historical MBS (reported at screening) as rows, and the MBS reported at the onset of the treated migraine as columns. This tabulation only includes subjects with both assessments. P-value from a chi-square test will be reported along with the values and confidence limits for both Asymmetric Lambda and Symmetric Lambda.

The estimand, difference in percentage of MBS free subjects ("risk difference") between treatment groups, is evaluated by computing the common risk difference, using CMH weights (sample size weights), stratified by the use of prophylactic migraine medication (yes or no). The risk difference will be tested at a two-sided alpha level of 0.05. Missing data at 2 hours post-dose will be imputed as failure (NC=F). Also, the use of rescue medication prior to providing data at the 2 hour assessment, taking IP prior to reporting the MBS, or failure to report a MBS are events that are imputed as treatment failures. If a stratum (prophylactic medication use: yes or no) has sparse data (less than 5 subjects) then the strata will be pooled.

The results to be presented for the primary analysis of MBS include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is now the probability of being MBS free at two-hours post-dose.

The primary analysis of MBS will be repeated for the subgroups described in Section 4.2.6.

Sensitivity analyses will be conducted as follows:

- 1. The primary analysis is repeated, using the mITT population, with missing data at 2 hours post-dose imputed using LOCF. BOCF is permitted.
- 2. The primary analysis is repeated, using only data from complete cases (data present at baseline and 2 hours).
- 3. The primary analysis is executed using the mITT analysis set, and multiple imputation (with 20 imputations; m=20) methods to impute missing data at 2 hours post-dose using the copy from reference approach. The FCS method is used with a generalized logit distribution. Covariates may include use of prophylactic medication (yes or no), sex, migraine intensity at onset (severe or other), migraines per month (< median, ≥ median), and the subject's MBS at time of study migraine onset (nausea, photophobia, or phonophobia).
- 4. A matrix of "what if" analyses, similar to that created for the co-primary endpoint of pain freedom, is created for freedom from the MBS.
- 5. The primary analysis will be repeated, using the mITT population, with the addition of a stratum that reflects the subject's self-reported MBS at the time of study migraine onset (nausea, phonophobia, or photophobia).

# 4.7.4 Secondary Efficacy Endpoints

If the co-primary endpoint tests are both significant, then the secondary endpoints are evaluated using a fixed sequence approach, with each test in the hierarchy conducted at p=0.05. See Section 4.2.5 for the testing order.

## 4.7.4.1 Freedom from Photophobia, Phonophobia or Nausea at 2 Hours

Freedom from photophobia, phonophobia, and nausea are assessed, by treatment group, by tabulating the number of mITT subjects who reported the presence of the symptom at migraine onset who then report the absence of the symptom at 2 hours post-dose. Subjects who report the symptom at baseline, but have missing data at 2 hours post-dose will be imputed as failures (NC=F). Also, subjects in the analysis set that take rescue medications on or before providing their 2 hours post-dose data are imputed as failures.

The principal measurement for the associated symptoms (phonophobia, photophobia, and nausea) is made on a binary scale (0 = absent; 1 = present). An exploratory measurement of these symptoms was also made on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).

For these three endpoints, the difference between treatment groups is evaluated by computing the common risk difference, using CMH weights (sample size weights), stratified by the use of prophylactic migraine medication (yes or no). The risk difference is tested at a two-sided alpha level of 0.05. If a stratum (prophylactic medication use: yes or no) has sparse data (less than 5 subjects) then the strata are pooled.

The results presented for the analysis of each symptom include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of being free from the symptom of interest at 2 hours post-dose. In addition, the following display will be created for each of the 3 symptoms:

A table showing descriptive statistics for the 4-point scale, which includes the number and percentage of subjects reporting each of the 4 symptom levels at 2 hours post-dose, and the percentage of subjects with missing data, for each treatment group. The table will include exact (Clopper-Pearson) 95% CIs for each percentage.

## 4.7.4.2 Pain Relief (at 60 Minutes; at 90 Minutes; at 2 Hours)

Pain relief at the specified timepoint post-dose is assessed by tabulating the number of mITT subjects that report a pain level of none or mild (responses of 0 or 1 on the 4-point Likert scale) at the specified timepoint post-dose, by treatment group. Subjects with missing data at the specified timepoint post-dose will be imputed as failures (NC=F).

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of pain relief at the specified timepoint post-dose.

## 4.7.4.3 Probability of Requiring Rescue Medication within 24 Hours

Whether or not a subject took rescue medication within 24 hours after the initial dose of study medication is tabulated by treatment group using mITT subjects, and the percentages are compared between treatment groups.

The results are presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of not requiring rescue medication within 24 hours post-dose.

Information regarding the rescue medication, including the type, date and time taken, dose, route and form of administration, and frequency, is presented in a listing by subject and treatment group.

# 4.7.4.4 Functional Disability Scale (at 60 Minutes; at 90 Minutes; at 2 Hours)

Impact of treatment on subject disability is assessed using a single-question, FDS. Subjects rate the level of disability they perceive as a result of their migraine in performing normal actions using a 4-point scale: Normal Function, Mild Impairment, Severe Impairment, or Required Bedrest. The proportion of mITT subjects who have a response of "normal" at the specified timepoint post dose will be evaluated as the endpoint of interest.

The information from the 4-point scale will be directly summarized as follows:

A table showing descriptive statistics for the 4-point scale, which includes the number and percentage of subjects reporting each of the 4 disability levels at the specified timepoint post-dose, and the percentage of subjects with missing data, for each treatment group, using the observed data. The table will include exact (Clopper-Pearson) 95% CIs for each percentage.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is now the probability of a functional disability level of "normal" at the specified timepoint post-dose.

### 4.7.4.5 Sustained Pain Freedom from 2 to 24 Hours

Sustained pain freedom is assessed using the number of mITT subjects that experienced no headache pain (response of 0 on Likert scale) at all time points from 2 through 24 hours post-dose. Subjects with missing pain scores at 1 or fewer time points, given that they have responses of no pain (response of 0 on 4-point Likert scale) at all other time points including the 2 and 24 hour post-dose time points, will be considered as successes. Subjects with responses missing at greater than 1 post-dose time point, missing data at the 2 or 24 hour time point, or with any pain score greater than 0 will be considered as failures.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained pain freedom from 2 to 24 hours.

#### 4.7.4.6 Sustained Pain Freedom from 2 to 48 Hours

Sustained pain freedom is assessed using the number of mITT subjects that experienced no headache pain (response of 0 on Likert scale) at all time points from 2 through 48 hours post-dose. Subjects with missing pain scores at no more than 1 time point, given that they have responses of no pain (response of 0 on Likert scale) at the 2, 24, and 48 hour time points will be considered as successes. Subjects with responses missing at greater than 1 time point; missing data at the 2, 24, or 48 hour time point; or with any pain score greater than 0 will be considered as failures

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained pain freedom from 2 to 48 hours.

### 4.7.4.7 Sustained Pain Relief from 2 to 24 Hours

Sustained pain relief is assessed using the number of mITT subjects who experience no or mild headache pain (responses of either 0 or 1 on 4-point Likert scale) at all time points from 2 through 24 hours post-dose. Subjects with missing pain scores at no more than 1 time point, given that they have responses of no or mild pain at the 2 and 24 hour time points will be considered as successes. Subjects with responses missing at more than 1 time point, with missing data at the 2 or 24 hour time points, or with any pain score greater than 1 will be considered as failures.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained pain relief from 2 to 24 hours.

#### 4.7.4.8 Sustained Pain Relief from 2 to 48 Hours

Sustained pain relief will be assessed using the number of subjects that experience no or mild headache pain (response of 0 or 1 on the 4-point Likert scale) at all time points from 2 through 48 hours post-dose. Subjects with missing pain scores at no more than 1 time point, given that they have responses of no or mild pain at all other time points including the 2, 24, and 48 hour time points will be considered as successes. Subjects with responses missing at more than 1 time point; with missing data at the 2, 24, or 48 hour time point; or with any pain score greater than 1 will be considered as failures

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained pain relief from 2 to 48 hours.

#### 4.7.4.9 Sustained MBS Freedom from 2 to 24 Hours

Sustained MBS freedom is assessed using the number of mITT subjects that experienced freedom from their MBS at all time points from 2 through 24 hours post-dose. Subjects with missing MBS scores at 1 or fewer time points, given that they have responses of freedom from

MBS at all other time points including the 2 and 24 hour post-dose time points will be considered as successes. Subjects with responses missing at greater than 1 post-dose time point, missing data at the 2 or 24 hour time point, or with any report of presence of MBS will be considered as failures.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained MBS freedom from 2 to 24 hours.

#### 4.7.4.10 Sustained MBS Freedom from 2 to 48 Hours

Sustained MBS freedom is assessed using the number of mITT subjects that experienced freedom from their MBS at all time points from 2 through 48 hours post-dose. Subjects with missing MBS scores at 1 or fewer time points, given that they have responses of freedom from MBS at all other time points including the 2, 24, and 48 hour post-dose time points will be considered as successes. Subjects with responses missing at greater than 1 post-dose time point, missing data at the 2, 24, or 48 hour time point, or with any report of presence of MBS will be considered as failures.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained MBS freedom from 2 to 48 hours.

# 4.7.4.11 Sustained Normal Functioning from 2 to 24 Hours

Sustained normal functioning is assessed using the number of mITT subjects that experienced normal functioning on the FDS at all time points from 2 through 24 hours post-dose. Subjects with missing FDS scores at 1 or fewer time points, given that they have responses of normal at all other time points including the 2 and 24 hour post-dose time points will be considered as successes. Subjects with responses missing at greater than 1 post-dose time point, missing data at the 2 or 24 hour time point, or with any report of non-normal functioning will be considered as failures.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained normal functioning from 2 to 24 hours.

### 4.7.4.12 Sustained Normal Functioning from 2 to 48 Hours

Sustained normal functioning is assessed using the number of mITT subjects that experienced normal functioning on the FDS at all time points from 2 through 48 hours post-dose. Subjects with missing FDS scores at 1 or fewer time points, given that they have responses of normal at all other time points including the 2, 24, and 48 hour post-dose time points will be considered as successes. Subjects with responses missing at greater than 1 post-dose time point, missing data at the 2, 24, or 48 hour time point, or with any report of non-normal functioning will be considered as failures.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained normal functioning from 2 to 48 hours.

#### 4.7.4.13 Pain Freedom at 90 Minutes

Pain freedom at 90 minutes post-dose is assessed by tabulating the number of mITT subjects that report a pain level of none (response of 0 on the 4-point Likert scale) at 90 minutes post-dose, by treatment group. Subjects with missing data at 90 minutes post-dose will be imputed as failures (NC=F).

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of pain freedom at 90 minutes post-dose.

#### 4.7.4.14 MBS Freedom at 90 Minutes

MBS freedom at 90 minutes post-dose is assessed by tabulating the number of mITT subjects that report an absence of their MBS at 90 minutes post-dose, by treatment group. Subjects with missing data at 90 minutes post-dose will be imputed as failures (NC=F).

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of MBS freedom at 90 minutes post-dose.

## 4.7.4.15 Pain Relapse from 2 to 48 Hours

Pain relapse is assessed using the number of mITT subjects that are pain free at 2 hours post-dose as the denominator. The numerator is the number of these subjects that then have a relapse of pain at any severity (response of 1, 2, or 3 on the 4-point Likert scale) within 48 hours after administration of study medication. Subjects with more than 1 time point with missing data or with missing data at the 2, 24, or 48 hour time point are classified as relapsers.

The results to be presented for the analysis include those described in items (a) through (e) for the primary analysis of pain freedom (Section 4.7.3.1). In this case, the "risk" is the probability of sustained pain relapse from 2 to 48 hours.

## 4.7.5 Exploratory Efficacy Endpoints

Any p-values presented for exploratory efficacy endpoints are for descriptive purposes only.

## 4.7.5.1 Functional Disability Scale at 24 Hours

Data will be analyzed in the same manner as described in Section 4.7.4.4. However, in this case the analysis will use the data from the 24 hour post-dose time point.

#### 4.7.5.2 Pain Relief at 15, 30, 60 and 90 Minutes Post-Dose

Pain relief at 15, 30, 60, and 90 minutes post-dose will be assessed by tabulating the number of mITT subjects that report a pain level of none or mild (responses of 0 or 1 on the 4-point Likert scale) at the specified post-dose time point by treatment group. Subjects with missing data at the specified post-dose time point will be imputed as failures (NC=F).

First, the data will be evaluated at each time point for each time point, using the first analysis methods described in Section 4.7.3.1.

Pain relief over time up to 8 hours will be analyzed using Kaplan-Meier methods. Kaplan-Meier estimates will be tabulated using the following time periods (0 through 15 minutes, >15 through 30 minutes, > 30 through 60 minutes, > 60 through 90 minutes, > 90 through 120 minutes, >120 minutes through 180 minutes, >180 minutes though 240 minutes, >240 minutes though 360 minutes, >360 minutes though 495 minutes, and > 495 minutes). For each time period, the number of subjects at risk, with an event (pain freedom), censored, and survival probability estimate (with 95% CI), will be presented by treatment group. Subjects who fail to reach no pain by 495 minutes, will be censored at 496 minutes. Additionally, subjects who take rescue medication prior to 495 minutes will be censored at the date/time associated with their rescue medication. Note that the probability of survival corresponds to the probability of NOT having pain relief. Survival estimates are calculated using the Kaplan-Meier product-limit method and median survival (time to pain freedom), and will be presented along with 95% CIs calculated using the method of Brookmeyer and Crowley.

To support the analysis, a Kaplan-Meier plot, with time in minutes on the x-axis and probability of survival on the y-axis, will be presented by treatment group. The number at risk at each time point (0, 15, 30, 45, 60, 90, 120, 180, 240, 360, and 495) minutes will be presented below the figure. In this analysis, being at risk corresponds to not yet having achieved pain relief; therefore, the subject is still "at risk" of having pain freedom. Once a subject has pain relief or is censored, then the subject is no longer in the risk pool. If a subject has missing data at an earlier time point, then the time point with missing data is not considered. The subject is still considered at risk of failure at a future time point if data are available. Subjects are censored as described above.

### 4.7.5.3 Preference of Medication (PoM)

The PoM is a brief scale that captures the subjects' perception of whether the medication they are taking has had a greater benefit compared with previous medications to treat their pain. Responses at 24 hours post-dose for all subjects who provided a response, and answered "yes" to the lead-in question (i.e. "Have you ever taken migraine medication"), will be tabulated. The number and percentage of subjects preferring the study medication, along with 95% asymptotic CIs, are presented by treatment group. The tabulations will be repeated for the subset of subjects considered as responders or non-responders by treatment group without imputation, where responders are those subjects who reported a pain score of 0 or 1 at 2 hours post-dose and who did not require rescue medication at or prior to 2 hours post-dose.

## 4.7.5.4 Migraine Quality of Life Questionnaire (MQoLQ)

Impact of treatment on patient-reported quality of life is assessed using the MQoLQ, which is a 15-item instrument that has been validated in migraine patients to measure the short-term impact of treatment (within 24 hours). The MQoLQ consists of 15 items across the following five domains: (1) work functioning, (2) social functioning, (3) energy/vitality, (4) migraine symptoms, and (5) feelings/concerns. There are three items within each domain. Response options for each of the items are on a 7-point scale where 1 indicates maximum impairment of QoL and 7 indicates no impairment. Each domain has a maximum score of 21 and a minimum score of 3. The items in the work functioning domain are: (1) ability to do normal everyday work, (2) ability to operate machinery or a motor vehicle, and (3) ability to stay alert. The items in the social functioning domain are: (1) interactions with people who are close to you, (2) interactions with other people, and (3) ability to enjoy life. The items in the energy/vitality domain are: (1) energy level, (2) ability to have a good night's sleep, and (3) mood. The items in the migraine symptoms domain are: (1) have throbbing head pain, (2) have increased sensitivity to light and/or noise, and (3) have nausea. Lastly, the items in the feelings/concerns domain are: (1) feel upset about having migraine headaches, (2) feel physically uncomfortable, and (3) feel concern that your migraine medication wouldn't relieve your migraine headache symptoms.

The observed responses at 24 hours post-dose will be presented for each item, each domain, and as a total score, by treatment group. The observed responses at 24 hours will also be summarized as a continuous response for each item, domain, and for the total score. Responses will also be presented in a by-subject listing along with treatment group, historical MBS collected at screening, MBS reported at migraine onset, migraine severity just prior to study medication, and migraine severity at 24 hours post-dose.

### 4.7.5.5 Efficacy at Each Pose-Dose Time Point

Pain freedom, pain relief, freedom from MBS, and functional disability score will be tabulated by treatment group at each post-dose time point. Success for each of these endpoints will be tabulated using the mITT subjects.

Freedom from nausea, freedom from phonophobia, freedom from photophobia, and FDS response will be tabulated by treatment group at each post-dose time point. The tabulation will include: the total number of subjects reporting each of the above symptoms at baseline, success as the percentage of the total number of subjects reporting the symptoms at baseline, and the number of subjects that reported the symptom but with missing data at the post-dose time point as a percentage of the number reporting the symptom at baseline.

#### 4.7.5.6 Pain Freedom to 8 Hours Post-Dose

Pain freedom over time up to 8 hours will be analyzed using Kaplan-Meier methods. Kaplan-Meier estimates will be tabulated using the following time periods (0 through 15 minutes, >15 through 30 minutes, > 30 through 60 minutes, > 60 through 90 minutes, > 90 through 120 minutes, >120 minutes through 180 minutes, >180 minutes though 240 minutes, >240 minutes though 360 minutes, >360 minutes though 495 minutes, and > 495 minutes). For each time period, the number of subjects at risk, with an event (pain freedom), censored, and survival
probability estimate (with 95% CI), will be presented by treatment group. Subjects who fail to reach no pain by 495 minutes, will be censored at 496 minutes. Additionally, subjects who take rescue medication prior to 495 minutes will be censored at the date/time associated with their rescue medication. Note that the probability of survival corresponds to the probability of NOT having pain freedom. Survival estimates are calculated using the Kaplan-Meier product-limit method and median survival (time to pain freedom), and will be presented along with 95% CIs calculated using the method of Brookmeyer and Crowley.

To support the analysis, a Kaplan-Meier plot, with time in minutes on the x-axis and probability of survival on the y-axis, will be presented by treatment group. The number at risk at each time point (0, 15, 30, 45, 60, 90, 120, 180, 240, 360, and 495) minutes will be presented below the figure. In this analysis, being at risk corresponds to not yet having achieved pain freedom; therefore, the subject is still "at risk" of having pain freedom. Once a subject has pain freedom or is censored, then the subject is no longer in the risk pool. If a subject has missing data at an earlier time point, then the time point with missing data is not considered. The subject is still considered at risk of failure at a future time point if data are available. Subjects are censored as described above.

#### 4.8 Pharmacokinetic Evaluation

No pharmacokinetic data will be collected in this study.

### 4.9 Safety Evaluation

Safety analyses will be conducted on the treated population by as-treated treatment group (i.e., the actual treatment received) and overall. All safety data will be presented in by-subject listings and will indicate which values are on-study or on-treatment.

Safety outcome measures include: AEs, laboratory assessments including liver toxicity, vital signs, physical measurements, electrocardiograms (ECGs), concomitant and rescue medications, and suicidal ideation and behaviors. Unless otherwise noted, baseline is considered as last non-missing assessment on or prior to study drug randomization.

### 4.9.1 Extent of Exposure

Extent of exposure is measured by subjects providing self-reported study drug exposure information in their eDiaries. As a check on this exposure data, study drug accountability data are provided by the study center on the "Drug Accountability" CRF page.

The self-reported study drug exposure data will be tabulated by treatment group and overall for randomized subjects who had an on-study migraine, and will include:

- The number (and percentage) of randomized subjects that took study medication
  - The number and percentage who took the medication prior to providing baseline study migraine characteristics

- The number and percentage that took study medication after providing baseline study migraine characteristics
- The number and percentage of randomized subjects who reported not taking study medication
- The number and percentage of randomized subjects for whom no exposure data was reported

The study drug accountability will be tabulated by treatment group and overall for randomized subjects who had an on-study migraine, and will include:

- The number and percentage of randomized subjects to whom kits were dispensed
- The number and percentage of kits returned
  - o The number and percentage of kits returned from which the IP was used
  - o The number and percentage of kits returned from which the IP was not used
- The number and percentage of kits not returned

A cross tabulation of exposure and accountability data will be prepared. This will be done overall for randomized subjects who had an on-study migraine. For the exposure and accountability data, the categories are: Took IP, Did not Take IP, and Unknown.

A by-subject listing will be prepared that indicates the study drug exposure and accountability status of all randomized subjects. A patient identifier (PID) listing will be prepared if subjects had unknown exposure data, unknown accountability data, or for whom the exposure and accountability data did not match.

#### 4.9.2 Adverse Events

AEs will be coded using MedDRA and displayed in tables and listings by SOC and PT, unless specified otherwise.

On-study AEs are those with a start (onset) date on or after the randomization date.

Adverse events are summarized by subject incidence rates; therefore, in any tabulation, a subject contributes only once to the count for a given AE (SOC or PT). The number and percentage of subjects with any on-study AE, with any on-study AE related to treatment (unlikely related, possibly related, or related), with any on-study SAE, with any on-study SAE related to treatment, with any on-study severe AE, with any on-study AE leading to study drug discontinuation and with any on-study AE leading to death will be summarized by treatment group and overall.

The number and percentage of subjects with on-study AEs will also be summarized by SOC and PT for the following: any AE; AEs related to study drug; SAEs; severe AEs; and AEs leading to study drug discontinuation. AEs will be displayed in descending order of overall frequency within SOC and PT.

In these tabulations, each subject will contribute only once (i.e., the most related occurrence or the most intense occurrence) to each of the incidence rates in the descriptive analysis, regardless of the number of episodes. All AEs will be listed and indicate whether or not the AE was serious, occurred on study, or potentially occurred on treatment. Additional listings will be provided including: deaths; SAEs; and AEs leading to study drug discontinuation.

Potentially on-treatment AEs are those with a start date on or after the first dose of study drug date. Given that the AEs do not have recorded onset times, these on-study events are considered to be potentially on-treatment. (Thus, potentially on-treatment AEs are a subset of on-study AEs).

### 4.9.3 Laboratory Data

Clinical laboratory evaluations include:

Hematology: hemoglobin, hematocrit, red blood cell count, white blood cell count with differential, and platelets

Serum Chemistry: sodium, potassium, chloride, bicarbonate, calcium, glucose, BUN (urea), serum creatinine, uric acid, ALT, AST, alkaline phosphatase, LDH, total protein, albumin, total bilirubin, direct bilirubin, indirect bilirubin, CPK (with fractionation, if available)

Lipid Panel: Cholesterol, LDL, HDL, triglycerides (screening only)

Estimated glomerular filtration rate (eGFR) using the estimated modification of diet in renal disease (MDRD) formula will be calculated and reported by the central lab at each visit that the clinical laboratory test is collected.

Urinalysis: pH, specific gravity, protein, ketones, nitrites, urobilinogen, leukocyte esterase, protein, glucose, microalbuminuria, and blood. If blood, protein, or leukocytes are positive, reflex to microscopic examination.

Urine drug screen: for drugs of abuse

Clinical laboratory values will be expressed using both Standard US units and SI units. Tabulations, listings, and graphics will be provided to show the data in both systems, unless specified otherwise.

The observed value and change from baseline will be summarized for select continuous laboratory parameters at baseline and the end of treatment visit. In addition, the shift from baseline in laboratory tests will be summarized as the number and percentage of subjects with each category (low, normal, high) at baseline and the end of treatment visit. Note that shift

categories are independent of US and SI units. For AST and ALT, the shift tables will use the following categories (SI and US units are the same): Normal, >ULN, >3x ULN, and >5x ULN. In the event of repeat values from the same post-baseline visit, the non-missing value closest to the target date for the visit will be used. In the case of a tie, the latest record will be used.

All laboratory data will be provided in by-subject listings that indicate which values are on study or on treatment. Additional listings will be presented for all abnormal laboratory values.

On-study laboratory values are those with collection date/time after the randomization date/time.

On-treatment laboratory values are those with collection date/time after the first dose of study drug date/time. (Thus, on-treatment laboratory values are a subset of on-study values.)

These definitions of on-study/on-treatment apply to vital signs, physical measurements, ECGs, and suicidal ideation and behaviors.

### 4.9.3.1 Liver Toxicity Evaluation

Potential drug induced liver injury (DILI) are those events meeting Hy's Law, defined as:

- 1. Aminotransferases (AT) ALT or AST elevation > 3 times the upper limit of normal (ULN);
- 2. Total bilirubin (TBL) > 2 times ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase); and
- 3. No other immediately apparent possible causes of AT elevation and hyperbilirubinemia, included but not limited to: viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic.

Any on-study potential DILI, meeting the above defined criteria, will be reported as SAEs in the SAE summary table (see Section 4.9.2). A by-subject listing of potential DILI will be prepared that shows the AT and TBL values for all subjects that experience either AT > 3 times the upper limit of normal or TBL > 2 times the upper limit of normal at any time.

Additionally, a table will be created that summarizes the on-study incidence (as the number and percentage of subjects with an elevation) of the following:

- >3x, >5x, >10x, and >20x ULN elevations of AST, ALT, and either ALT or AST
- Any elevations of bilirubin >1x ULN and >2x ULN
- Any elevations of ALP > 1.5x ULN
- Elevation of AST or ALT (>3x ULN) accompanied by elevated bilirubin (>1.5x ULN and >2x ULN)

• Elevation of AST or ALT along with an on-study AE of nausea, vomiting, anorexia, abdominal pain, or fatigue

An evaluation of on-study Drug-Induced Serious Hepatotoxicity (eDISH) plot will be created by plotting the maximum total bilirubin against maximum ALT and presenting these data points by treatment group. The maximum values for each subject during the study will be identified as the maximum values that occur on study, but not necessarily concurrently. Maximum total bilirubin (presented as xULN) will be plotted on a log scale on the y-axis and maximum ALT (presented as xULN) will be plotted on a log scale on the x-axis. A horizontal reference line will be placed at 2x ULN for maximum total bilirubin, and a vertical reference line will be placed at 3x ULN for maximum ALT. The lower left quadrant will be labeled "Normal Range". The upper left quadrant will be labeled "Hyperbilirubinemia". The lower right quadrant will be labeled "Possible Hy's Law Range".

### 4.9.4 Vital Signs and Physical Measurements

The observed value and change from baseline in vital signs will be summarized at baseline and the end of treatment visit.

### 4.9.5 Electrocardiogram

The shift from baseline in ECG parameters will be summarized as the number and percentage of subjects with normal and abnormal results at baseline and the end of treatment visit. The observed value and change from baseline in ECG interval data (e.g., RR, QRS, PR, QT, QTcF), and ventricular heart rate will also be summarized at baseline and the end of treatment visit.

### 4.9.6 Non-Study Medications

Concomitant medications will be coded using the WHO-DD. Results will be tabulated by Anatomic Therapeutic Class (ATC) and PT in descending order of overall frequency. For each subject, multiple records of the same medication will be counted only once within each ATC and/or PT.

The following non-study medications will be tabulated:

- Prior medications, defined as non-study medications with start or stop date < randomization date 14 days.
- Concomitant medications, defined as non-study medications with start or stop date ≥ randomization date − 14 days.
- Prophylactic medications taken at or after informed consent and before randomization, defined as those with (1) informed consent date ≤ start or stop date < randomization date, or (2) start date ≤ informed consent date and randomization date − 1 day ≤ stop date

- Prophylactic medications taken at or after randomization, defined as those with start or stop date ≥ randomization date.
- Rescue medications (see Section 4.7.1).

### 4.9.7 Sheehan-Suicidality Tracking Scale (S-STS)

The S-STS is a prospective, self-reported rating scale that contains 16 questions to track both treatment-emergent suicidal ideation and behaviors. In the event the subject is unavailable, the S-STS clinician-administered rating scale will be completed that contains 6 yes/no questions.

Self-reported S-STS scores are calculated as follows:

Ideation subscale score: Sum of scores (0-4) for Questions 2-11

Behavior subscale score: Sum of scores (0-4) for Questions 1a, (highest of 12 or any row of 16), (highest of 14 or any row of 15), 17, and 20

Total score: Sum of the ideation and behavior subscale scores

The self-reported S-STS ideation subscale, behavior subscale, and total score will be summarized at baseline, and the number and percentage of subjects in change from baseline categories (i.e., <-1, -1, no change, 1, >1) will be summarized at the end of treatment visit.

# APPENDIX 1: TABLES, LISTINGS, AND FIGURES

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.1.1 | Subject Disposition | Enrolled Subjects | Y |
| 14.1.2.1 | Demographic and Baseline Characteristics | mITT Subjects | Y |
| 14.1.2.2 | Demographic and Baseline Characteristics | Subjects Enrolled but Not Randomized | |
| 14.1.2.3 | Demographic and Baseline Characteristics | Subjects Randomized but Not Treated | |
| 14.1.2.4 | Demographic and Baseline Characteristics | Treated Subjects | |
| 14.1.3.1 | Medical History by System Organ Class and Preferred Term | mITT Subjects | |
| 14.1.3.2 | Medical History by System Organ Class and Preferred Term | Treated Subjects | |
| 14.1.4.1 | Migraine History | mITT Subjects | Y |
| 14.1.4.2 | Migraine History | Subjects Enrolled but Not Randomized | |
| 14.1.4.3 | Migraine History | Subjects Randomized but Not Treated | |
| 14.1.4.4 | Migraine History | Treated Subjects | |
| 14.1.5.1 | Cardiac and Other Risk Factors | mITT Subjects | |
| 14.1.5.2 | Cardiac and Other Risk Factors | Treated Subjects | |
| 14.1.6.1 | Prior Triptan Response | mITT Subjects | |
| 14.1.6.2 | Prior Triptan Response | Treated Subjects | |
| 14.1.7.1 | Current Triptan Response | mITT Subjects | |
| 14.1.7.2 | Current Triptan Response | Treated Subjects | |
| 14.1.8 | Subgroup Summary | mITT Subjects | Y |
| 14.1.9.1 | Missing Data Summary for Primary and Secondary Efficacy Endpoints | Randomized Subjects | |
| 14.1.9.2 | Missing Pain Data at 2 Hours Post Dose Summary by Subgroup | mITT Subjects | |
| 14.2.1.1.1 | Pain Freedom at 2 Hours Post Dose: Observed Data | mITT Subjects | |
| 14.2.1.1.1.2 | Pain Freedom at 2 Hours Post Dose: Asian Subjects Only | mITT Subjects | |
| 14.2.1.1.2 | Pain Freedom at 2 Hours Post Dose: Primary Analysis | mITT Subjects | Y |
| 14.2.1.1.3.1 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by Age | mITT Subjects | |
| 14.2.1.1.3.2 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by Race | mITT Subjects | |
| 14.2.1.1.3.3 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by Sex | mITT Subjects | |
| 14.2.1.1.3.4 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by Aura | mITT Subjects | |
| 14.2.1.1.3.5 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by Headaches | mITT Subjects | |
| | per Month | | |
| 14.2.1.1.3.6 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by Prior Triptan | mITT Subjects | |
| | Response | | |
| 14.2.1.1.3.7 | Pain Freedom at 2 Hours Post Dose: Subgroup Analysis by | mITT Subjects | |
| | Cardiovascular Risk | | |

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.1.1.4.1 | Pain Freedom at 2 Hours Post Dose: Sensitivity Analysis 1: Applying Last Observation Carried Forward | mITT Subjects | |
| 14.2.1.1.4.2 | Pain Freedom at 2 Hours Post Dose: Sensitivity Analysis 2: Complete Case Analysis | mITT Subjects | |
| 14.2.1.1.4.3 | Pain Freedom at 2 Hours Post Dose: Sensitivity Analysis 3: Multiple Imputation | mITT Subjects | |
| 14.2.1.1.4.4 | Pain Freedom at 2 Hours Post Dose: Sensitivity Analysis 4: Varying Success Rate Imputations | mITT Subjects | |
| 14.2.1.1.4.5 | Pain Freedom at 2 Hours Post Dose: Sensitivity Analysis 5: Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.1.2 | Most Bothersome Symptom at Migraine Onset: Observed Data | mITT Subjects | |
| 14.2.1.2.1.1 | Historically Most Bothersome Symptom versus Most Bothersome<br>Symptom at Migraine Onset | mITT Subjects | |
| 14.2.1.2.1.2 | Most Bothersome Symptom Score at 2 Hours Post Dose: Observed Data | mITT Subjects | |
| 14.2.1.2.2 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Primary Analysis | mITT Subjects | Y |
| 14.2.1.2.3.1 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Age | mITT Subjects | |
| 14.2.1.2.3.2 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Race | mITT Subjects | |
| 14.2.1.2.3.3 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Sex | mITT Subjects | |
| 14.2.1.2.3.4 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Aura | mITT Subjects | |
| 14.2.1.2.3.5 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Headaches per Month | mITT Subjects | |
| 14.2.1.2.3.6 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Prior Triptan Response | mITT Subjects | |
| 14.2.1.2.3.7 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Subgroup Analysis by Cardiovascular Risk | mITT Subjects | |
| 14.2.1.2.4.1 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Sensitivity Analysis 1: Applying Last Observation Carried Forward | mITT Subjects | |
| 14.2.1.2.4.2 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Sensitivity Analysis 2: Complete Case Analysis | mITT Subjects | |
| 14.2.1.2.4.3 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Sensitivity Analysis 3: Multiple Imputation | mITT Subjects | |
| 14.2.1.2.4.4 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Sensitivity Analysis 4: Varying Success Rate Imputations | mITT Subjects | |

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.1.2.4.5 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Sensitivity Analysis 5: Stratified by MBS at Study Migraine Onset | mITT Subjects | |
| 14.2.1.2.4.6 | Freedom from Most Bothersome Symptom at 2 Hours Post Dose:<br>Sensitivity Analysis 6: Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.1.1 | Freedom from Photophobia at 2 Hours Post Dose in Subjects who Reported Photophobia at Study Migraine Onset: Observed Data | mITT Subjects | |
| 14.2.2.1.2 | Freedom from Photophobia at 2 Hours Post Dose in Subjects who Reported Photophobia at Study Migraine Onset: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.1.3 | Freedom from Photophobia at 2 Hours Post Dose in Subjects who<br>Reported Photophobia at Study Migraine Onset: Secondary Analysis<br>Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.2.1 | Freedom from Phonophobia at 2 Hours Post Dose in Subjects who Reported Phonophobia at Study Migraine Onset: Observed Data | mITT Subjects | |
| 14.2.2.2.2 | Freedom from Phonophobia at 2 Hours Post Dose in Subjects who Reported Phonophobia at Study Migraine Onset: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.2.3 | Freedom from Phonophobia at 2 Hours Post Dose in Subjects who<br>Reported Phonophobia at Study Migraine Onset: Secondary Analysis<br>Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.3.1 | Freedom from Nausea at 2 Hours Post Dose in Subjects who Reported Nausea at Study Migraine Onset: Observed Data | mITT Subjects | |
| 14.2.2.3.2 | Freedom from Nausea at 2 Hours Post Dose in Subjects who Reported Nausea at Study Migraine Onset: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.3.3 | Freedom from Nausea at 2 Hours Post Dose in Subjects who Reported Nausea at Study Migraine Onset: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.4.1 | Pain Relief at 60 Minutes Post Dose: Observed Data | mITT Subjects | |
| 14.2.2.4.2 | Pain Relief at 60 Minutes Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.4.3 | Pain Relief at 60 Minutes Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.5.1 | Pain Relief at 90 Minutes Post Dose: Observed Data | mITT Subjects | |
| 14.2.2.5.2 | Pain Relief at 90 Minutes Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.5.3 | Pain Relief at 90 Minutes Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.6.1 | Pain Relief at 2 Hours Post Dose: Observed Data | mITT Subjects | |
| 14.2.2.6.2 | Pain Relief at 2 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.6.3 | Pain Relief at 2 Hours Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.7.1 | Rescue Medication within 24 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.2.7.2 | Rescue Medication within 24 Hours Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.8.1 | Functional Disability Scale at 60 Minutes Post Dose: Observed Data | mITT Subjects | |
| 14.2.2.8.2 | Functional Disability Scale at 60 Minutes Post Dose: Secondary Analysis mITT Subjects | | |
| 14.2.2.8.3 | Functional Disability Scale at 60 Minutes Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.9.1 | Functional Disability Scale at 90 Minutes Post Dose: Observed Data | mITT Subjects | |
| 14.2.2.9.2 | Functional Disability Scale at 90 Minutes Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.9.3 | Functional Disability Scale at 90 Minutes Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.10.1 | Functional Disability Scale at 2 Hours Post Dose: Observed Data | mITT Subjects | |
| 14.2.2.10.2 | Functional Disability Scale at 2 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.10.3 | Functional Disability Scale at 2 Hours Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.11.1 | Sustained Pain Freedom from 2 to 24 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.11.2 | Sustained Pain Freedom from 2 to 48 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.11.3 | Sustained Pain Relief from 2 to 24 Hours Post Dose: Secondary<br>Analysis | mITT Subjects | Y |
| 14.2.2.11.4 | Sustained Pain Relief from 2 to 48 Hours Post Dose: Secondary<br>Analysis | mITT Subjects | Y |
| 14.2.2.11.5 | Sustained Pain Freedom from 2 to 24 Hours Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.11.6 | Sustained Pain Freedom from 2 to 48 Hours Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.11.7 | Sustained Pain Relief from 2 to 24 Hours Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.11.8 | Sustained Pain Relief from 2 to 48 Hours Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.12.1 | Sustained MBS Freedom from 2 to 24 Hours Post Dose: Secondary Analysis | | |
| 14.2.2.12.2 | Sustained MBS Freedom from 2 to 48 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.12.3 | Sustained MBS Freedom from 2 to 24 Hours Post Dose: Secondary<br>Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.2.12.4 | Sustained MBS Freedom from 2 to 48 Hours Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.13.1 | Sustained Normal Functioning from 2 to 24 Hours Post Dose:<br>Secondary Analysis | mITT Subjects | Y |
| 14.2.2.13.2 | Sustained Normal Functioning from 2 to 48 Hours Post Dose: mITT Subjects Secondary Analysis | | |
| 14.2.2.13.3 | Sustained Normal Functioning from 2 to 24 Hours Post Dose:<br>Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.13.4 | Sustained Normal Functioning from 2 to 48 Hours Post Dose:<br>Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.14.1 | Pain Freedom at 90 Minutes Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.14.2 | Pain Freedom at 90 Minutes Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.15.1 | Freedom from Most Bothersome Symptom at 90 Minutes Post Dose:<br>Secondary Analysis | mITT Subjects | Y |
| 14.2.2.15.2 | Freedom from Most Bothersome Symptom at 90 Minutes Post Dose:<br>Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.2.16.1 | Pain Relapse from 2 to 48 Hours Post Dose: Secondary Analysis | mITT Subjects | Y |
| 14.2.2.16.2 | Pain Relapse from 2 to 48 Hours Post Dose: Secondary Analysis Excluding Site 002 | mITT Subjects Excluding Site 002 | |
| 14.2.3.1 | Functional Disability Scale at 24 Hours Post Dose: Exploratory Analysis | mITT Subjects | |
| 14.2.3.2 | Pain Relief at 15 and 30 Minutes Post Dose: Exploratory Analysis | mITT Subjects | |
| 14.2.3.3.1 | Kaplan-Meier Time to First Report of Pain Relief up to 8 Hours Post Dose: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.3.2 | Median Time to First Report of Pain Relief: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.4 | Preference of Medication at 24 Hours Post Dose: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.5.1 | Migraine Quality of Life Questionnaire at 24 Hours Post Dose:<br>Continuous Exploratory Analysis | mITT Subjects | |
| 14.2.3.5.2 | Migraine Quality of Life Questionnaire at 24 Hours Post Dose:<br>Frequency Exploratory Analysis | mITT Subjects | |
| 14.2.3.6 | Pain Freedom at Every Timepoint Post Dose: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.7 | Pain Relief at Every Timepoint Post Dose: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.8 | Freedom from Most Bothersome Symptom at Every Timepoint Post<br>Dose: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.9 | Freedom from Photophobia at Every Timepoint Post Dose: Exploratory Analysis | mITT Subjects | |
| 14.2.3.10 | Freedom from Phonophobia at Every Timepoint Post Dose: Exploratory Analysis | mITT Subjects | |

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.3.11 | Freedom from Nausea at Every Timepoint Post Dose: Exploratory Analysis | mITT Subjects | |
| 14.2.3.12 | Functional Disability Scale at Every Timepoint Post Dose: Exploratory Analysis | mITT Subjects | Y |
| 14.2.3.13.1 | Kaplan-Meier Time to First Report of Pain Freedom up to 8 Hours Post Dose: Exploratory Analysis | Kaplan-Meier Time to First Report of Pain Freedom up to 8 Hours Post | |
| 14.2.3.13.2 | Median Time to First Report Pain Freedom: Exploratory Analysis | mITT Subjects | Y |
| 14.3.1.1 | Self-Reported Study Drug Exposure Summary | All Randomized Subjects who had a Study Migraine | |
| 14.3.1.2 | Study Drug Accountability Summary | All Randomized Subjects who had a Study Migraine | |
| 14.3.1.3 | Cross Tabulation of Study Drug Exposure and Accountability | All Randomized Subjects who had a Study Migraine | |
| 14.3.2.1 | Summary of On-Study Adverse Events | Treated Subjects | Y |
| 14.3.2.2 | Incidence of On-study Adverse Events by System Organ Class and Preferred Term | Treated Subjects | Y |
| 14.3.2.3 | Incidence of On-study Adverse Events Related to Study Drug by System Organ Class and Preferred Term | Treated Subjects | |
| 14.3.2.4 | Incidence of On-study Serious Adverse Events by System Organ Class and Preferred Term | Treated Subjects | Y |
| 14.3.2.5 | Incidence of On-study Adverse Events with Severe Grade by System Organ Class and Preferred Term | Treated Subjects | Y |
| 14.3.2.6 | Incidence of On-Study Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term | Treated Subjects | |
| 14.4.1.1 | Hematology (SI Units): Observed and Change From Baseline Values by Visit | Treated Subjects | |
| 14.4.1.2 | Hematology (UI Units): Observed and Change From Baseline Values by Visit | Treated Subjects | |
| 14.4.2.1 | Serum Chemistry (SI Units): Observed and Change From Baseline<br>Values by Visit | Treated Subjects | |
| 14.4.2.2 | Serum Chemistry (US Units): Observed and Change From Baseline<br>Values by Visit | Treated Subjects | |
| 14.4.3 | Hematology: Shift from Baseline by Visit | Treated Subjects | |
| 14.4.4 | Serum Chemistry: Shift from Baseline by Visit | Treated Subjects | |
| 14.4.5 | Urinalysis: Shift from Baseline by Visit | Treated Subjects | |
| 14.4.5.2 | Urine Drug Screen: Shift from Baseline by Visit | Treated Subjects | |
| 14.4.6 | Transaminases: Shift from Baseline by Visit | Treated Subjects | |
| 14.4.7 | Summary of On-Study Liver Toxicity | Treated Subjects | Y |

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.5.1 | Vital Signs and Physical Measurements: Observed and Change from | Treated Subjects | |
| | Baseline Values by Visit | | |
| 14.5.2.1 | Electrocardiogram: Observed and Change from Baseline Values by Visit | Treated Subjects | |
| 14.5.2.2 | Electrocardiogram: Shift from Baseline by Visit | Treated Subjects | |
| 14.5.3.1 | Prior Non-Study Medications by Therapeutic Class and Preferred Term | Treated Subjects | |
| 14.5.3.2 | Concomitant Non-Study Medications by Therapeutic Class and | Treated Subjects | |
| | Preferred Term | | |
| 14.5.3.3 | Non-Study Prophylactic Migraine Medications Taken at or After | Treated Subjects | |
| | Informed Consent and Before Randomization by Therapeutic Class and | | Y |
| | Preferred Term | | |
| 14.5.3.4 | Non-Study Prophylactic Migraine Medications Taken at or After | Treated Subjects | v |
| | Randomization by Therapeutic Class and Preferred Term | | 1 |
| 14.5.3.5 | Non-Study Rescue Medicationsby Therapeutic Class and Preferred | Treated Subjects | v |
| | Term | | I |
| 14.5.4 | Sheehan-Suicidality Tracking Scale: Exploratory Analysis | Treated Subjects | |

| <b>Listing Number</b> | Title | Population | Topline |
|---|---|---|---|
| 16.2.1.1 | Subject Disposition | Enrolled Subjects | |
| 16.2.1.2 | Subject Eligibility | Enrolled Subjects | |
| 16.2.1.3 | Significant Protocol Deviations | Enrolled Subjects | |
| 16.2.2.1 | Demographic and Baseline Characteristics | Enrolled Subjects | |
| 16.2.2.2 | Medical History | Enrolled Subjects | |
| 16.2.2.3 | General Migraine History | Enrolled Subjects | |
| 16.2.2.4 | Migraine Symptom History | Enrolled Subjects | |
| 16.2.2.5 | Migraine Aura Symptom History | Enrolled Subjects | |
| 16.2.2.6 | Cardiac and Other Risk Factors | Enrolled Subjects | |
| 16.2.2.7 | Reasons for Discontinuation from Prior Triptans | Enrolled Subjects | |
| 16.2.2.8 | Current Triptan Response | Enrolled Subjects | |
| 16.2.3 | Batch Numbers | Enrolled Subjects | |
| 16.2.4 | Subpopulations and Subgroups | mITT Subjects | |
| 16.2.5.1 | Observed Pain and MBS Efficacy Measurements | mITT Subjects | |
| 16.2.5.2 | Observed Primary Efficacy Measurements at 2 Hours Post Dose | mITT Subjects | |
| 16.2.5.3 | Functional Disability Scale | mITT Subjects | |
| 16.2.5.4 | Preference of Medication at 24 Hours Post Dose | mITT Subjects | |
| 16.2.5.5 | Migraine Quality of Life Questionnaire at 24 Hours Post Dose | mITT Subjects | |
| 16.2.6 | Study Drug Exposure and Accountability | Randomized Subjects | |

| 16.2.7.1 | Adverse Events | Enrolled Subjects |
|---|---|---|
| 16.2.7.2 | Serious Adverse Events | Enrolled Subjects |
| 16.2.7.3 | Deaths | Enrolled Subjects |
| 16.2.7.4 | Adverse Events Leading to Study Drug Discontinuation | Treated Subjects |
| 16.2.8.1.1 | Hematology Results (SI Units) | Enrolled Subjects |
| 16.2.8.1.2 | Hematology Results (US Units) | Enrolled Subjects |
| 16.2.8.2.1 | Serum Chemistry Results (SI Units) | Enrolled Subjects |
| 16.2.8.2.2 | Serum Chemistry Results (US Units) | Enrolled Subjects |
| 16.2.8.2.3 | CK and Fractionation Results (SI Units) | Enrolled Subjects |
| 16.2.8.2.4 | CK and Fractionation Results (US Units) | Enrolled Subjects |
| 16.2.8.3.1 | Urinalysis Results (SI Units) | Enrolled Subjects |
| 16.2.8.3.2 | Urinalysis Results (US Units) | Enrolled Subjects |
| 16.2.8.3.3 | Urine Drug Screen Results | Enrolled Subjects |
| 16.2.8.4.1 | Endocrine Results (SI Units) | Enrolled Subjects |
| 16.2.8.4.2 | Endocrine Results (US Units) | Enrolled Subjects |
| 16.2.8.5.1 | Pregnancy Test Results (SI Units) | Enrolled Subjects |
| 16.2.8.5.2 | Pregnancy Test Results (US Units) | Enrolled Subjects |
| 16.2.8.6 | GC/MS Results | Enrolled Subjects |
| 16.2.8.7.1 | All Abnormal Laboratory Results (SI Units) | Enrolled Subjects |
| 16.2.8.7.2 | All Abnormal Laboratory Results (US Units) | Enrolled Subjects |
| 16.2.8.8.1 | Potential Drug Induced Liver Injury (SI Units) | Enrolled Subjects |
| 16.2.8.8.2 | Potential Drug Induced Liver Injury (US Units) | Enrolled Subjects |
| 16.2.9.1 | Vital Signs and Physical Measurements | Enrolled Subjects |
| 16.2.9.2 | Electrocardiogram Results | Enrolled Subjects |
| 16.2.9.3.1 | Non-Study Medications | Enrolled Subjects |
| 16.2.9.3.2 | Non-Study Prophylactic Migraine Medications | Enrolled Subjects |
| 16.2.9.3.3 | Rescue Medications | Enrolled Subjects |
| 16.2.9.4 | Procedures | Enrolled Subjects |
| 16.2.9.5 | Sheehan-Suicidality Tracking Scale Results | Enrolled Subjects |

| Figure Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.1 | Forest Plot of Pain Freedom at 2 Hours Post Dose | mITT Subjects | |
| 14.2.1.1 | Forest Plot of Pain Freedom at 2 Hours Post Dose: Sensitivity | mITT Subjects | |
| | Analysis 1 | | |

| 14.2.1.2 | Forest Plot of Pain Freedom at 2 Hours Post Dose: Sensitivity<br>Analysis 2 | mITT Subjects | |
|---|---|---|---|
| 14.2.1.3 | Forest Plot of Pain Freedom at 2 Hours Post Dose: Sensitivity<br>Analysis 3 | mITT Subjects | |
| 14.2.1.4 | Forest Plot of Pain Freedom at 2 Hours Post Dose: Sensitivity<br>Analysis 4 | mITT Subjects | |
| 14.2.1.5 | Forest Plot of Pain Freedom at 2 Hours Post Dose by Subgroup | mITT Subjects | |
| 14.2.2 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose | mITT Subjects | |
| 14.2.2.1 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose: Sensitivity Analysis 1 | mITT Subjects | |
| 14.2.2.2 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose: Sensitivity Analysis 2 | mITT Subjects | |
| 14.2.2.3 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose: Sensitivity Analysis 3 | mITT Subjects | |
| 14.2.2.4 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose: Sensitivity Analysis 4 | mITT Subjects | |
| 14.2.2.5 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose: Sensitivity Analysis 5 | mITT Subjects | |
| 14.2.2.6 | Forest Plot of Freedom from Most Bothersome Symptom at 2 Hours<br>Post Dose by Subgroup | mITT Subjects | |
| 14.2.3 | Forest Plot of Freedom from Photophobia, Phonophobia, and Nausea at 2 Hours Post Dose | mITT Subjects | |
| 14.2.4 | Forest Plot of Pain Relief | mITT Subjects | |
| 14.2.5 | Forest Plot of Probability of Requiring Rescue Medication within 24 Hour Post Dose | mITT Subjects | |
| 14.2.6 | Forest Plot of Probability of Functioning Normally According to the Functional Disability Scale | mITT Subjects | |
| 14.2.7.1 | Forest Plot of Durability of Pain Relief | mITT Subjects | |
| 14.2.7.2 | Forest Plot of Durability of Pain Freedom | mITT Subjects | |
| 14.2.7.3 | Forest Plot of Durability of MBS Freedom | mITT Subjects | |
| 14.2.7.4 | Forest Plot of Durability of Normal Functioning | mITT Subjects | |
| 14.2.7.5 | Forest Plot of Probability of Pain Relapse | mITT Subjects | |
| 14.2.8 | Kaplan-Meier Plot of Time to First Report of Pain Relief up to Eight Hours Post Dose | mITT Subjects | Y |
| 14.2.9 | Kaplan-Meier Plot of Time to First Report of Pain Freedom to Eight Hours Post Dose | mITT Subjects | Y |
| 14.3.1 | Evaluation of On-Study Drug-Induced Hepatotoxicity (eDISH) | Treated Subjects | Y |

# APPENDIX 2: SCHEDULE OF ASSESSMENTS

| <u>Procedure</u> | Screening Visit (3-28 days) | Baseline Visit<br>(Randomization) <sup>1</sup> | Onset of<br>moderate or<br>severe<br>migraine <sup>2</sup> | During Treatment 15, 30, 45, 60 and 90 minutes Post-Dose | During Treatment 2, 3, 4, 6, 8 hours Post- Dose | During Treatment 24 hours Post-Dose | During Treatment 48 hours Post- Dose | End of<br>Treatment<br>Visit |
|---|---|---|---|---|---|---|---|---|
| Eligibility Assessments | | | | | | | | |
| Informed Consent | X | | | | | | | |
| Inclusion/Exclusion<br>Criteria | х | X | | | | | | |
| Medical History | X | | | | | | | |
| Prophylactic Migraine<br>Medication/ Concomitant<br>Medication <sup>3</sup> | x | х | | | | | | х |
| Assessment of Migraine<br>History (Signs and<br>symptoms) paper<br>source <sup>14</sup> | х | | | | | | | |
| Safety Assessments | | | | | | | | |
| Physical Examination | X | | | | | | | X |
| Vital Signs/Physical<br>Measurements <sup>4</sup> | x | x | | | | | | х |
| Clinical Safety<br>Laboratory Testing <sup>5</sup> | X | | | | | | | х |

| <u>Procedure</u> | Screening Visit (3-28 days) | Baseline Visit<br>(Randomization) <sup>1</sup> | Onset of<br>moderate or<br>severe<br>migraine <sup>2</sup> | During Treatment 15, 30, 45, 60 and 90 minutes Post-Dose | During Treatment 2, 3, 4, 6, 8 hours Post- Dose | During<br>Treatment<br>24 hours<br>Post-Dose | During Treatment 48 hours Post- Dose | End of<br>Treatment<br>Visit |
|---|---|---|---|---|---|---|---|---|
| ECG | X | | | | | | | X |
| Pregnancy Test <sup>6</sup> | х | Х | х | | | | | х |
| Adverse Event and<br>Serious Adverse Event<br>Assessment <sup>7</sup> | х | х | x | x | х | х | x | х |
| Sheehan Suicidality<br>Tracking Scale <sup>8</sup> | Х | Х | | | | | | X |
| Clinical Drug<br>Supplies/Study Supplies | | | | | | | | |
| Randomize <sup>9</sup> | | X | | | | | | |
| Dispense Study<br>Medication | | X | | | | | | |
| Administer 1 dose of<br>study medication <sup>10</sup> | | | х | | | | | |
| Return unused study<br>medication | | | | | | | | Х |
| eDiary returned/reviewed<br>for completeness <sup>11</sup> | | | | | | | | х |
| Efficacy Assessments <sup>12</sup> | | | | | | | | |
| Assessment of migraine pain 13 | | | х | х | х | х | x | |

| <u>Procedure</u> | Screening Visit (3-28 days) | Baseline Visit<br>(Randomization) <sup>1</sup> | Onset of<br>moderate or<br>severe<br>migraine <sup>2</sup> | During Treatment 15, 30, 45, 60 and 90 minutes Post-Dose | During Treatment 2, 3, 4, 6, 8 hours Post- Dose | During<br>Treatment<br>24 hours<br>Post-Dose | During<br>Treatment<br>48 hours<br>Post- Dose | End of<br>Treatment<br>Visit |
|---|---|---|---|---|---|---|---|---|
| Assessment of Migraine<br>Symptoms (photophobia,<br>phonophobia, and nausea<br>- eDiary) <sup>13</sup> | | | х | х | х | х | х | |
| Functional Disability<br>Scale <sup>13</sup> | | | X | X | X | X | Х | |
| MQoLQ (Migraine<br>Specified Quality of Life<br>Questionnaire) <sup>13</sup> | | | | | | x | | |
| Preference of<br>Medication <sup>13</sup> | | | | | | x | | |

<sup>&</sup>lt;sup>1</sup> Screening/Baseline Phase will be 3 - 28 days. The Baseline Visit may be scheduled but should only occur *after* all screening procedures are complete, patient meets inclusion/exclusion criteria, and lab test results have been received by the site.

<sup>&</sup>lt;sup>2</sup> Patients will use eDiary to answer questions about their migraine symptoms upon experiencing a moderate/severe migraine headache. The patient will administer predispensed study drug if 1) the headache remains moderate or severe; 2) the patient has completed all required migraine assessment questions in the eDiary, including their current most bothersome migraine symptom, and 3) the patient has not already taken prohibited medications (see protocol section 5.4).

<sup>&</sup>lt;sup>3</sup> Patients should keep track of their concomitant medications throughout the study and report them to the study personnel at the End of Treatment Visit. Any medication taken for recurrent headache should be documented. Use of concomitant medications after randomization, including rescue medications, will be recorded by the patient on a paper diary and reported to the site.

<sup>&</sup>lt;sup>4</sup> Height will only be captured at the Screening Visit. Weight body temperature, respiratory rate, blood pressure and heart rate will be collected at all time points where indicated. Sitting arterial systolic and diastolic blood pressure and pulse rate will be measured.

<sup>&</sup>lt;sup>5</sup> All Screening Visit laboratory test results must be received prior to Baseline Visit.

<sup>&</sup>lt;sup>6</sup> A serum pregnancy test will be completed at Screening and End of Treatment Visits as part of the standard laboratory tests (if appropriate). Confirmatory urine pregnancy test for WOCBP should be completed on site at Baseline Visit and any subsequent visits for confirmation at the Investigator's discretion. Home pregnancy test will be provided to WOCBP after completion of baseline visit.

<sup>&</sup>lt;sup>7</sup> SAEs are reported from the time of informed consent and non-serious AEs are reported from baseline. All ongoing non-serious AEs and SAEs will be followed to resolution or until investigator deems there will be no further status change. SAE and AE's that occur during the treatment period should be reported to the site.

<sup>&</sup>lt;sup>8</sup> This scale will be clinician administered, completed on site, and will be in paper. The source document will be provided by Biohaven. The assessment period for completing the scale will be 30 days prior to Screening, and since the last visit for the remainder of the study.

<sup>&</sup>lt;sup>9</sup> Patients will be randomized in the IWRS system at the Baseline Visit (Randomization Day 01)

<sup>&</sup>lt;sup>10</sup> Patient should be instructed that the dose should be taken once the migraine attack reaches moderate or severe pain.

<sup>&</sup>lt;sup>11</sup> Site staff to review and confirm entries with patients and confirm all data points are transferred to the system and reset eDiary for future patient use, PRIOR to the patient leaving the clinic.

<sup>&</sup>lt;sup>12</sup> ± Windows for timeframe around efficacy assessments (15, 30, 45, 60, 90 min, 2, 3, 4, 6, 8, 24 and 48 hours) will be automated and captured in the eDiary.

<sup>13</sup> These scales will be captured in the eDiary. Patients will also be asked about their most bothersome symptom at the time of reporting and treating a qualifying migraine.

<sup>14</sup> Paper source document will be used to capture Migraine History. Patients will also be asked about their typical most bothersome symptom when having a migraine.

### **APPENDIX 3: SUPPORTIVE ANALYSES**

### 1 DURABILITY ENDPOINTS

New durability endpoints were defined for pain freedom, pain relief, most bothersome symptom, functional disability, nausea, photophobia, and phonophobia. For each of these endpoints, durability was measured during six time periods:

- 2 to 24 hours
- 3 to 24 hours
- 4 to 24 hours
- 2 to 48 hours
- 3 to 48 hours
- 4 to 48 hours

For pain freedom and pain relief, the 2 to 24 hour and 2 to 48 hour durability endpoints were previously defined in the SAP in Sections 5.7.4.5 - 5.7.4.8.

Pain freedom, pain relief, most bothersome symptom, and functional disability were assessed using the mITT population. Nausea, photophobia, and phonophobia were assessed using mITT subjects who reported the given symptom as present at the start of their treated migraine.

For all ad-hoc durability endpoints, the following were presented:

- The number and percentage of subjects who are successful. These are presented by stratum and treatment group, with ASE and 95% asymptotic CIs.
- Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.
- Risk difference within each strata with sample size, p-value, ASE and 95% asymptotic CIs.
- A plot of the risk differences within each strata, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

The "risk" is the probability of the given endpoint (success) through the given durability period.

### 1.1 Sustained Pain Freedom

The ad-hoc sustained pain freedom endpoints were:

- Sustained Pain Freedom 3 to 24 hours
- Sustained Pain Freedom 4 to 24 hours
- Sustained Pain Freedom 3 to 48 hours
- Sustained Pain Freedom 4 to 48 hours

Sustained pain freedom for the above time periods were defined in a manner similar to that used for sustained pain freedom from 2 to 24 hours and 2 to 48 hours.

Sustained pain freedom was assessed using the number of mITT subjects who experienced no headache pain (response of 0 on the Likert scale) at all time points from the starting time point (3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing pain scores at 1 or fewer time points, given that they had responses of no pain at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any pain score greater than 0 were considered as failures.

### 1.2 Sustained Pain Relief

The ad-hoc sustained pain relief endpoints were:

- Sustained Pain Relief 3 to 24 hours
- Sustained Pain Relief 4 to 24 hours
- Sustained Pain Relief 3 to 48 hours
- Sustained Pain Relief 4 to 48 hours

Sustained pain relief for the above time periods were defined in a manner similar to that used previously for sustained pain relief from 2 to 24 hours and 2 to 48 hours.

Sustained pain relief was assessed using the number of mITT subjects who experienced no or mild headache pain (response of 0 or 1 on the Likert scale) at all time points from the starting time point (3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing pain scores at 1 or fewer time points, given that they had responses of no or mild pain at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any pain score greater than 1 were considered as failures.

## 1.3 Sustained Freedom from Most Bothersome Symptom

The ad-hoc sustained freedom from the MBS endpoints were:

- Sustained Freedom from MBS 2 to 24 hours
- Sustained Freedom from MBS 3 to 24 hours
- Sustained Freedom from MBS 4 to 24 hours
- Sustained Freedom from MBS 2 to 48 hours
- Sustained Freedom from MBS 3 to 48 hours
- Sustained Freedom from MBS 4 to 48 hours

Sustained freedom from MBS for these time periods is defined in a manner similar to that used for sustained pain freedom from 2 to 24 hours and 2 to 48 hours.

Sustained MBS freedom was assessed using the number of mITT subjects who did not have their MBS (response of absent) at all time points from the starting time point (2, 3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing MBS scores at 1 or fewer time points, given that they had responses of absent MBS at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any MBS present at any time point in the period were considered as failures.

### 1.4 Sustained Freedom from Functional Disability

The ad-hoc sustained freedom from functional disability endpoints were:

- Sustained Freedom from Functional Disability 2 to 24 hours
- Sustained Freedom from Functional Disability 3 to 24 hours
- Sustained Freedom from Functional Disability 4 to 24 hours
- Sustained Freedom from Functional Disability 2 to 48 hours
- Sustained Freedom from Functional Disability 3 to 48 hours
- Sustained Freedom from Functional Disability 4 to 48 hours

Sustained freedom from functional disability for these time periods is defined in a manner similar to that used for sustained pain freedom from 2 to 24 hours and 2 to 48 hours.

Sustained freedom from functional disability was assessed using the number of mITT subjects who experienced normal functioning at all time points from the starting time point (2, 3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing disability scores at 1 or fewer time points, given that they have responses of no disability at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any reported disability in the time period were classified as failures.

#### 1.5 Sustained Freedom from Nausea

The ad-hoc sustained freedom from nausea endpoints were:

- Sustained Freedom from Nausea 2 to 24 hours
- Sustained Freedom from Nausea 3 to 24 hours
- Sustained Freedom from Nausea 4 to 24 hours
- Sustained Freedom from Nausea 2 to 48 hours
- Sustained Freedom from Nausea 3 to 48 hours
- Sustained Freedom from Nausea 4 to 48 hours

Sustained freedom from nausea for these time periods was defined in a manner similar to that used for sustained pain freedom from 2 to 24 hours and 2 to 48 hours. However, the analysis population was restricted to those subjects with nausea reported as present at the start of their treated migraine.

Sustained nausea freedom was assessed using the number of mITT subjects who had nausea present at baseline and did not report nausea (response of absent) at any time point from the starting time point (2, 3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing nausea scores at 1 or fewer time points, given that they had responses of no nausea at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any nausea present at any time point in the period were considered as failures.

### 1.6 Sustained Freedom from Photophobia

The ad-hoc sustained freedom from photophobia endpoints are:

- Sustained Freedom from Photophobia 2 to 24 hours
- Sustained Freedom from Photophobia 3 to 24 hours
- Sustained Freedom from Photophobia 4 to 24 hours
- Sustained Freedom from Photophobia 2 to 48 hours
- Sustained Freedom from Photophobia 3 to 48 hours
- Sustained Freedom from Photophobia 4 to 48 hours

Sustained freedom from photophobia for these time periods was defined in a manner similar to that used for sustained freedom from nausea. The analysis population was restricted to those mITT subjects with photophobia reported as present at the start of their treated migraine.

Sustained photophobia freedom was assessed using the number of mITT subjects who had photophobia present at baseline and that did not report photophobia (response of absent) at any time point from the starting time point (2, 3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing photophobia scores at 1 or fewer time points, given that they had responses of no photophobia at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any photophobia present at any time point in the period were considered as failures.

### 1.7 Sustained Freedom from Phonophobia

The ad-hoc sustained freedom from phonophobia endpoints are:

- Sustained Freedom from Phonophobia 2 to 24 hours
- Sustained Freedom from Phonophobia 3 to 24 hours
- Sustained Freedom from Phonophobia 4 to 24 hours
- Sustained Freedom from Phonophobia 2 to 48 hours
- Sustained Freedom from Phonophobia 3 to 48 hours
- Sustained Freedom from Phonophobia 4 to 48 hours

Sustained freedom from phonophobia for these time periods was defined in a manner similar to that used for sustained freedom from nausea. The analysis population was restricted to those mITT subjects with phonophobia reported as present at the start of their treated migraine.

Sustained phonophobia freedom was assessed using the number of mITT subjects who had phonophobia present at baseline and that did not report phonophobia (response of absent) at any time point from the starting time point (2, 3 or 4 hours post-dose) through the ending time point (24 or 48 hours post-dose). Subjects with missing phonophobia scores at 1 or fewer time points, given that they had responses of no phonophobia at all other time points including the starting and ending time points (and 24 hours for periods through 48 hours), were considered as successes. Subjects with missing data at greater than 1 post-dose time point, missing data at either the starting or ending time point (or 24 hours for periods through 48 hours), or with any phonophobia present at any time point in the period were considered as failures.

### 2 TIME TO EVENT ANALYSES

#### 2.1 Time to Rescue Medication

Kaplan-Meier plots were created for the time to first use of rescue medication. The K-M plot covered the 24 hour period after dosing. Subjects who did not take rescue medication within 24 hours of dosing were censored at 24 hours and 1 minute. Regardless of pain or MBS response, subjects were considered at risk until the first use of rescue medication, loss to follow-up (last contact date), or the end of the 24 hour period, whichever came first. The analysis population consisted of mITT subjects.

Two tables were created to support the plot. The first table presented the median time to rescue medication along with 95% CIs calculated using the method of Brookmeyer and Crowley and the log-rank p-value. The second table presented the number of subjects at risk, with an event, censored, and the survival probability estimate (with 95% CI) for each period by treatment group.

### 2.2 Time to First Report of Absence of Various Symptoms

For each of the following variables, two sets of Kaplan-Meier plots and tables were created:

- Time to First Report of Absence of Most Bothersome Symptom
- Time to First Report of Absence of Nausea
- Time to First Report of Absence of Photophobia
- Time to First Report of Absence of Phonophobia
- Time to First Report of Return to Normal Functioning

The first set of plots and tables was similar to those created for the time to rescue medication (using actual time). For the second set of plots, nominal (planned time point) as opposed to actual time was used for clinical event times. Censoring was measured using actual time as in all previous plots.

For both sets of analyses, the analysis population for MBS was the set of mITT subjects. The analysis population for nausea, phonophobia, and photophobia was the subset of mITT subjects that reported the symptom as present at the onset of their study migraine. The analysis population for functional disability was the subset of mITT subjects that reported abnormal functioning at the onset of their study migraine. The y-axis for all plots represents the probability of the occurrence of the event of interest, and therefore are increasing from left to right.

### 2.2.1 Kaplan-Meier Plots and Tables: Actual Time for Event of Interest

The first set of K-M plots and tables were created using actual time of censoring and actual time for the clinical event of interest. Subjects were censored at the actual time of their first use of rescue medication or last reported data point if lost to follow-up. Subjects who did not have the clinical event of interest by 8 hours post dose were censored at 496 minutes (480 minutes + 15 minute window + 1 minute).

### 2.2.2 Kaplan-Meier Plots and Tables: Nominal Time for Event of Interest

The second set of K-M plots and tables were created for the above variables with nominal time (planned time of collection, e.g., 2 hours, 3 hours, etc.) used for clinical events of interest and actual time used for censoring events. Subjects were censored at the actual time of their first use of rescue medication or last reported data point if lost to follow-up. Subjects who did not have the clinical event of interest by 8 hours post dose were censored at 496 minutes (480 minutes + 15 minute window + 1 minute).

### 3 PAIN AND MBS AT 3 HOURS POST DOSE

#### 3.1 Pain Freedom at 3 Hours Post Dose

The between group difference in the percentage of subjects with pain freedom at 3 hours post-dose was assessed by computing the "risk difference" between treatment groups. This was evaluated by computing the common risk difference, using CMH weights (sample size weights), stratified by the use of prophylactic migraine medication (yes or no). The risk difference was tested at a two-sided alpha level of 0.05. Missing data at 2 hours post-dose were imputed as failures (NC=F).

Results presented for this analysis included the following:

- Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.
- Risk difference within each strata with sample size, p-value, ASE, and 95% asymptotic CIs.
- A plot of the risk differences within each strata, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

#### 3.2 Freedom from MBS at 3 Hours Post Dose

The estimand, difference in percentage of subjects with freedom from MBS at 3 hours between treatment groups was evaluated by computing the common risk difference using CMH weights (sample size weights), stratified by the use of prophylactic migraine medication (yes or no). The risk difference was tested at a two-sided alpha level of 0.05. Missing data at 3 hours post-dose was imputed as failure (NC=F). Also the use of rescue medication prior to providing data at the 3 hour assessment, taking IP prior to reporting the MBS, or failure to report a MBS are events that were imputed as treatment failures.

Results presented for this analysis included the following:

- Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.
- Risk difference within each strata with sample size, p-value, ASE, and 95% asymptotic CIs.
- A plot of the risk differences within each strata, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

### 4 OTHER ENDPOINTS AT 3 HOURS POST DOSE

### 4.1 Freedom from Photophobia, Phonophobia, or Nausea at 3 Hours

Freedom from photophobia, phonophobia, and nausea were assessed, by treatment group, by tabulating the number of mITT subjects who reported the presence of the symptom at migraine onset, and later reported the absence of the symptom at 3 hours post-dose. Subjects who reported the symptom at baseline, but have missing data at 3 hours post-dose were imputed as failures (NC=F). Also, subjects in the analysis set who took rescue medications on or before providing their 3 hour post-dose data were imputed as failures.

The principal measurement for the associated symptoms (phonophobia, photophobia, and nausea) is made on a binary scale (0 = absent; 1 = present). An exploratory measurement of these symptoms was also made on a 4-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).

For these three endpoints, the difference between treatment groups, was evaluated by computing the common risk difference using CMH weights (sample size weights), stratified by the use of prophylactic migraine medication (yes or no). The risk difference was tested at a two-sided alpha level of 0.05.

Results presented for these analyses included the following:

• Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.

- Risk difference within each strata with sample size, p-value, ASE, and 95% asymptotic CIs.
- A plot of the risk differences within each strata, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

#### 4.2 Pain Relief at 3 Hours Post Dose

Pain relief at 3 hours post-dose was assessed by tabulating the number of mITT subjects that reported a pain level of none or mild (responses of 0 or 1 on the 4-point Likert scale) at 3 hours post-dose by treatment group. Subjects with missing data at 3 hours post-dose were imputed as failures (NC=F). Also, subjects in the analysis set who took rescue medications on or before providing their 3 hour post-dose data were imputed as failures.

Results presented for this analysis included the following:

- Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.
- Risk difference within each strata with sample size, p-value, ASE, and 95% asymptotic CIs.
- A plot of the risk differences within each strata, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

### 4.3 Functional Disability Scale at 3 Hours Post Dose

Impact of treatment on subject disability was assessed using a single-question, functional disability scale. Subjects rated the level of disability they perceived as a result of their migraine in performing normal actions using a 4-point scale: Normal Function, Mild Impairment, Severe Impairment, or Required Bedrest. The proportion of mITT subjects who had a response of "normal" at 3-hours post dose was evaluated as the endpoint of interest.

Results presented for this analysis included the following:

- Common risk difference with sample size, p-value, ASE, and 95% asymptotic CIs.
- Risk difference within each strata with sample size, p-value, ASE, and 95% asymptotic CIs.
- A plot of the risk differences within each strata, and common risk difference (similar to the risk difference plot produced by SAS Proc Freq).
- Common risk for each treatment with sample size, ASE, and 95% asymptotic CIs.

# APPENDIX 4: TABLES AND FIGURES FOR SUPPORTIVE ANALYSES

| Table Number | Title | Population | Topline |
|---|---|---|---|
| 14.2.1.1.4.6 | Pain Freedom at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.1.2.4.7 | Freedom from Most Bothersome Symptom at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.1.4 | Freedom from Photophobia at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.2.2.4 | Freedom from Phonophobia at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.3.4 | Freedom from Nausea at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.6.4 | Pain Relief at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.7.3 | Kaplan-Meier Time to Rescue Medication up to 24 hours Post Dose: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.7.4 | Median Time to Rescue Medication: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.10.4 | Functional Disability Scale at 3 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.11.9 | Sustained Pain Freedom from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.11.10 | Sustained Pain Freedom from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.11.11 | Sustained Pain Relief from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.11.12 | Sustained Pain Relief from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.11.13 | Sustained Pain Freedom from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.11.14 | Sustained Pain Freedom from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.11.15 | Sustained Pain Relief from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.11.16 | Sustained Pain Relief from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.5 | Sustained MBS Freedom from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.6 | Sustained MBS Freedom from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.7 | Sustained MBS Freedom from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.8 | Sustained MBS Freedom from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.8.1 | Kaplan-Meier Time to First Report of Absence of MBS up to 8 hours Post Dose: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.12.8.2 | Median Time to First Report of Absence of MBS: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.12.8.3 | Kaplan-Meier Nominal Time to First Report of Absence of MBS up to 8 hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.8.4 | Median Nominal Time to First Report of Absence of MBS: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.9 | Sustained Nausea Freedom from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.10 | Sustained Nausea Freedom from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.11 | Sustained Nausea Freedom from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.12 | Sustained Nausea Freedom from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.13 | Sustained Photophobia Freedom from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.14 | Sustained Photophobia Freedom from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.15 | Sustained Photophobia Freedom from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.16 | Sustained Photophobia Freedom from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.17 | Sustained Phonophobia Freedom from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.18 | Sustained Phonophobia Freedom from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |

| 14.2.2.12.19 | Sustained Phonophobia Freedom from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
|---|---|---|---|
| 14.2.2.12.20 | Sustained Phonophobia Freedom from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.14.1 | Kaplan-Meier Time to First Report of Absence of Nausea up to 8 hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.14.2 | Median Time to First Report of Absence of Nausea: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.14.3 | Kaplan-Meier Nominal Time to First Report of Absence of Nausea up to 8 hours Post Dose: Ad-hoc | mITT Subjects | |
| | Analysis | , | |
| 14.2.2.12.14.4 | Median Nominal Time to First Report of Absence of Nausea: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.20.1 | Kaplan-Meier Time to First Report of Absence of Photophobia up to 8 hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.20.2 | Median Time to First Report of Absence of Photophobia: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.20.3 | Kaplan-Meier Nominal Time to First Report of Absence of Photophobia up to 8 hours Post Dose: Ad-hoc | mITT Subjects | |
| | Analysis | | |
| 14.2.2.12.20.4 | Median Nominal Time to First Report of Absence of Photophobia: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.26.1 | Kaplan-Meier Time to First Report of Absence of Phonophobia up to 8 hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.26.2 | Median Time to First Report of Absence of Photophobia: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.12.26.3 | Kaplan-Meier Nominal Time to First Report of Absence of Phonophobia up to 8 hours Post Dose: Ad-hoc | mITT Subjects | |
| | Analysis | | |
| 14.2.2.12.26.4 | Median Nominal Time to First Report of Absence of Photophobia: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.13.5 | Sustained Functional Disability Freedom from 3 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.13.6 | Sustained Functional Disability Freedom from 4 to 24 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.13.7 | Sustained Functional Disability Freedom from 3 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.13.8 | Sustained Functional Disability Freedom from 4 to 48 Hours Post Dose: Ad-hoc Analysis | mITT Subjects | |
| 14.2.2.13.8.1 | Kaplan-Meier Time to First Report of Return to Normal Functioning up to 8 hours Post Dose: Ad-hoc | mITT Subjects | Y |
| | Analysis | | - |
| 14.2.2.13.8.2 | Median Time to First Report of Return to Normal Functioning: Ad-hoc Analysis | mITT Subjects | Y |
| 14.2.2.13.8.3 | Kaplan-Meier Nominal Time to First Report of Return to Normal Functioning up to 8 hours Post Dose: Ad- | mITT Subjects | |
| | hoc Analysis | | |
| 14.2.2.13.8.4 | Median Nominal Time to First Report of Return to Normal Functioning: Ad-hoc Analysis | mITT Subjects | |

| Figure | Title | Population | Topline |
|---|---|---|---|
| Number | | | |
| 14.2.10 | Kaplan Meier Survival Plot of Time to Rescue Medication up to 24 Hours Post Dose | mITT Subjects | Y |
| 14.2.11 | Kaplan Meier Survival Plot of Time to First Report of Absence of MBS up to 8 Hours Post Dose | mITT Subjects | |
| 14.2.12 | Kaplan Meier Survival Plot of Time to First Report of Absence of Nausea up to 8 Hours Post Dose | mITT Subjects | |
| 14.2.13 | Kaplan Meier Survival Plot of Time to First Report of Absence of Photophobia up to 8 Hours Post Dose | mITT Subjects | |
| 14.2.14 | Kaplan Meier Survival Plot of Time to First Report of Absence of Phonophobia up to 8 Hours Post Dose | mITT Subjects | |
| 14.2.15 | Kaplan Meier Survival Plot of Time to First Report of Return to Normal Functioning up to 8 Hours Post | mITT Subjects | V |
| | Dose | | Y |

| 14.2.16 | Kaplan Meier Survival Plot of Time to First Report of Absence of MBS up to 8 Hours Post Dose (Nominal Time) | mITT Subjects | |
|---|---|---|---|
| 14.2.17 | Kaplan Meier Survival Plot of Time to First Report of Absence of Nausea up to 8 Hours Post Dose (Nominal Time) | mITT Subjects | |
| 14.2.18 | Kaplan Meier Survival Plot of Time to First Report of Absence of Photophobia up to 8 Hours Post Dose (Nominal Time) | mITT Subjects | |
| 14.2.19 | Kaplan Meier Survival Plot of Time to First Report of Absence of Phonophobia up to 8 Hours Post Dose (Nominal Time) | mITT Subjects | |
| 14.2.20 | Kaplan Meier Survival Plot of Time to First Report of Return to Normal Functioning up to 8 Hours Post Dose (Nominal Time) | mITT Subjects | Y |